CLINICAL TRIAL: NCT02203305
Title: Cochlear Implantation in Cases of Single-Sided Deafness
Acronym: CI in SSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-1544
Record Dates: First submitted 2014-07-22; First posted 2014-07-29 (Estimated); Results first posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-02

CONDITIONS: Unilateral Moderate to Profound Hearing Loss; Asymmetric Hearing Loss; Single-Sided Deafness (SSD)
Keywords: Unilateral hearing loss; Single Sided Deafness; Asymmetric hearing loss
MeSH Terms: conditions — Hearing Loss, Unilateral | interventions — Cochlear Implants; Control Groups

ARMS (3):
- Cochlear Implant (Experimental): Cochlear implantation of the affected ear
  Interventions: Device: Cochlear Implant
- Control Group (Other): A control group without the study intervention (cochlear implantation) will complete the test battery.
  Interventions: Other: Control Group
- Cochlear Implant: Asymmetric hearing loss (Experimental): Cochlear implantation of the poorer hearing ear
  Interventions: Device: Cochlear Implant

INTERVENTIONS:
Device: Cochlear Implant — cochlear implantation used a treatment for single-sided deafness and/or asymmetric hearing loss
  Other Names: MED-EL CONCERT cochlear implant system; MED-EL SYNCHRONY cochlear implant system
  Arms: Cochlear Implant; Cochlear Implant: Asymmetric hearing loss
Other: Control Group — Subjects in the control group will have had listening experience with a bone-conduction device, which is an approved treatment for SSD.
  Other Names: bone-conduction device
  Arms: Control Group

SUMMARY:
The primary goal of this project is to determine whether subjects with Single-Sided Deafness (SSD) experience an improvement in speech perception, localization, and quality of life with a cochlear implant as compared to an unaided listening condition.

DETAILED DESCRIPTION:
Single-sided deafness (SSD) can be defined as moderate-to-profound sensorineural hearing loss with limited speech perception benefit in one ear and normal hearing in the contralateral ear. Though one ear is within the normal hearing limits, SSD may result in reduced speech perception in noise, variable abilities on localization tasks, increased subjective report of hearing handicap, and reduced quality of life.

This patient population cannot utilize conventional amplification due to the severity of the hearing loss and poor speech discrimination abilities in the affected ear. Current treatment options include: contralateral routing of the signal (CROS) hearing aids, and bone-conduction devices. A CROS hearing aid is a two-part system that includes a microphone/transmitter on the affected ear and a receiver on the normal hearing ear. The microphone/transmitter sends the acoustic signal from the affected ear to the receiver, which is presented to the normal hearing ear. Bone-conduction devices utilize a percutaneous, implanted titanium abutment to send the acoustic signal from the affected side to the normal hearing ear via vibrations. The goal of both of these technologies is to send the signal from the affected side to the normal hearing side, thereby leaving the patient in a unilateral listening condition.

Though CROS hearing aids and bone-conduction devices provide the patient with auditory information from both sides to the better hearing ear, the ability to use binaural cues for speech perception in noise is variable.

It is of interest whether cochlear implantation of the affected ear would benefit the SSD population. A cochlear implant is a two-part system, including the internal electrode array and external speech processor. The internal electrode array is surgically implanted into the affected cochlea. The external speech processor receives sounds and transmits this signal to the internal portion. The electrode array presents the acoustic signal via electrical pulses within the cochlea, which is interpreted by the brain as sound.

Presumably, cochlear implantation may provide the SSD population improvements in speech perception in the affected ear, which cannot benefit from appropriately fit hearing aids. Cochlear implantation may provide a benefit over current treatment options in the SSD population, as it stimulates the auditory pathway on the affected side, thus allowing for ipsilateral representation of acoustic signals arriving to each ear independently.

The primary goal of this project is to determine whether subjects with SSD experience an improvement in speech perception, localization, and quality of life with a cochlear implant as compared to an unaided listening condition. Secondary aims include: 1) a comparison of speech perception, localization, and quality of life outcomes in the study population to a SSD control group with long-term listening experience with a current treatment option (i.e. bone-conduction device), and 2) a within-subject comparison of speech perception and localization abilities with cochlear implantation versus the bone-conduction test device.

ELIGIBILITY:
Inclusion Criteria (SSD):

* Unilateral moderate-to-profound sensorineural hearing loss [Unaided residual hearing thresholds measured from 250-8000 Hertz (Hz) (Pure Tone Average (PTA) ≥70 decibel (dB) Hearing Level (HL) in the ear to be implanted]
* Normal to mild residual hearing thresholds from 250-8000 Hz in the contralateral ear (≤35 dB HL at each frequency, 250-8000 Hz)
* Greater than or equal to 18 years of age at implantation
* Duration of moderate-to-profound sensorineural hearing loss less than or equal to 5 years [Either reported by subject or documented in previous audiograms] [Can be less than or equal to 10 years if the subject consistently utilized hearing technology (such as a bone conduction device or conventional hearing aid) within the past 5 years]
* Previous experience with a current treatment option for SSD, including a conventional hearing aid, bone-conduction device, or CROS/BICROS (Bilateral Contralateral Routing Of the Signal) technology. [At least one month of listening experience with device] [Dissatisfaction with and/or discontinued use of current treatment option due to: insufficient gain, poor sound quality, and/or lack of perceived benefit]
* Aided word recognition in the ear to be implanted of 60% or less as measured with Consonant-Nucleus-Consonant (CNC) words (50-word list) [When listening with an appropriately fit hearing aid and masking applied to the contralateral ear] [Aided testing will be conducted in a sound-proof booth with the subject seated 1 meter from the sound source, facing 0° azimuth. Recorded materials will be presented at 60 dB Sound Pressure Level (SPL).] [The hearing aid output will be measured using National Acoustic Laboratory-NonLinear (NAL-NL1) targets.]
* Realistic expectations
* Willing to obtain recommended meningitis vaccinations per Center for Disease Control (CDC) recommendations
* No reported cognitive issues [Pass the Mini Mental State Examination (MMSE) screener]
* Able and willing to comply with study requirements, including travel to investigational site and study-related activities

Exclusion Criteria (SSD):

* Non-native English speaker [Speech perception materials are presented in English]
* Conductive hearing loss in either ear
* Compromised auditory nerve, including those with a history of vestibular schwannoma
* Ossification
* Inability to participate in follow-up procedures (i.e., unwillingness, geographic location)
* History of meningitis, autoimmune disease, or any medical condition that contraindicate middle or inner ear surgery or anesthesia
* Meniere's disease with intractable vertigo
* Trauma that precludes inner ear surgery
* Case of sudden sensorineural hearing loss that has not been first evaluated by a physician
* Pregnancy [Subjects who are pregnant or become pregnant prior to surgery are excluded due to the potential risk of anesthesia to an unborn child.] [Subjects who become pregnant after surgery may continue to participate in study procedures]
* Tinnitus as the primary purpose for seeking cochlear implantation
* Subject obtains a severe or catastrophic score on the Tinnitus Handicap Inventory (Newman, Jacobson & Spitzer, 1996).

Inclusion Criteria (asymmetric hearing loss):

a. Ear to be implanted i. Moderate-to-profound sensorineural hearing loss ii. PTA ≥70 dB HL iii. Aided word recognition of 60% or less as measured with CNC words (50-word list).

b. Contralateral ear i. PTA ≥35 and ≤55 dB HL ii. Aided word recognition of 80% or more as measured with CNC words (50-word list).

iii. Use of conventional amplification c. Greater than or equal to 18 years of age at implantation d. Duration of moderate-to-profound sensorineural hearing loss in the ear to be implanted is less than or equal to 5 years [Either reported by subject or documented in previous audiograms. Can be up to 10 years if the subject consistently utilized hearing technology in the ear to be implanted (such as a bone conduction device or conventional hearing aid) within the past 5 years] e. Previous experience with a current treatment option for asymmetric hearing loss, including a conventional hearing aid, bone-conduction device, or CROS/BiCROS technology. [At least one month of listening experience with device. Dissatisfaction with and/or discontinued use of current treatment option due to: insufficient gain, poor sound quality, and/or lack of perceived benefit.] f. Realistic expectations g. Willing to obtain recommended meningitis vaccinations per CDC recommendations h. No reported cognitive issues [Pass the Mini Mental State Examination (MMSE) screener] i. Able and willing to comply with study requirements, including travel to investigational site and study-related activities

Exclusion Criteria (Asymmetric hearing loss):

1. Non-English speaker [Speech perception materials are presented in English]
2. Medical condition considered a contraindication to undergoing cochlear implantation
3. Conductive hearing loss in either ear
4. Compromised auditory nerve, including those with a history of vestibular schwannoma
5. Ossification
6. Inability to participate in follow-up procedures (i.e., unwillingness, geographic location)
7. History of meningitis, autoimmune disease, or any medical condition that contraindicate middle or inner ear surgery or anesthesia
8. Meniere's disease with intractable vertigo
9. Trauma that precludes inner ear surgery
10. Case of sudden sensorineural hearing loss that has not been first evaluated by a physician
11. Pregnancy [Subjects who are pregnant or become pregnant prior to surgery are excluded due to the potential risk of anesthesia to an unborn child. Subjects who become pregnant after surgery may continue to participate in study procedures]
12. Tinnitus as the primary purpose for seeking cochlear implantation
13. Subject obtains a severe or catastrophic score on the Tinnitus Handicap Inventory (Newman, Jacobson & Spitzer, 1996).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Dillon, AuD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Arndt S, Aschendorff A, Laszig R, Beck R, Schild C, Kroeger S, Ihorst G, Wesarg T. Comparison of pseudobinaural hearing to real binaural hearing rehabilitation after cochlear implantation in patients with unilateral deafness and tinnitus. Otol Neurotol. 2011 Jan;32(1):39-47. doi: 10.1097/MAO.0b013e3181fcf271. PMID 21068690
- [Background] Firszt JB, Holden LK, Reeder RM, Waltzman SB, Arndt S. Auditory abilities after cochlear implantation in adults with unilateral deafness: a pilot study. Otol Neurotol. 2012 Oct;33(8):1339-46. doi: 10.1097/MAO.0b013e318268d52d. PMID 22935813
- [Background] Hansen MR, Gantz BJ, Dunn C. Outcomes after cochlear implantation for patients with single-sided deafness, including those with recalcitrant Meniere's disease. Otol Neurotol. 2013 Dec;34(9):1681-7. doi: 10.1097/MAO.0000000000000102. PMID 24232066
- [Background] Vermeire K, Van de Heyning P. Binaural hearing after cochlear implantation in subjects with unilateral sensorineural deafness and tinnitus. Audiol Neurootol. 2009;14(3):163-71. doi: 10.1159/000171478. Epub 2008 Nov 13. PMID 19005250
- [Derived] Dillon MT, Buss E, Anderson ML, King ER, Deres EJ, Buchman CA, Brown KD, Pillsbury HC. Cochlear Implantation in Cases of Unilateral Hearing Loss: Initial Localization Abilities. Ear Hear. 2017 Sep/Oct;38(5):611-619. doi: 10.1097/AUD.0000000000000430. PMID 28375876

RESULTS

PARTICIPANT FLOW:
Groups:
- Cochlear Implant: Unilateral Hearing Loss Group: Cochlear implantation of the affected ear
  Cochlear Implant: cochlear implantation used a treatment for single-sided deafness and/or asymmetric hearing loss
- Cochlear Implant: Asymmetric Hearing Loss Group: Cochlear implantation of the poorer hearing ear
  Cochlear Implant: cochlear implantation used a treatment for single-sided deafness and/or asymmetric hearing loss
Period: Overall Study
Arm/Group | Cochlear Implant: Unilateral Hearing Loss Group | Control Group | Cochlear Implant: Asymmetric Hearing Loss Group
Started | 20 | 3 | 20
Completed | 20 | 3 | 19
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cochlear Implant: Unilateral Hearing Loss/Single-sided Deafness Group: Cochlear implantation of the affected ear
  Cochlear Implant: cochlear implantation used as a treatment for single-sided deafness/unilateral hearing loss and/or asymmetric hearing loss
- Cochlear Implant: Asymmetric Hearing Loss Group: Cochlear implantation of the poorer hearing ear
  Cochlear Implant: cochlear implantation used as a treatment for single-sided deafness/unilateral hearing loss and/or asymmetric hearing loss
- Total: Total of all reporting groups
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Deafness Group | Control Group | Cochlear Implant: Asymmetric Hearing Loss Group | Total
Number analyzed (Participants) | 20 | 3 | 20 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] — Age (years) at the time of cochlear implantation for treatment groups (unilateral hearing loss/single-sided deafness and asymmetric hearing loss). Age (years) at the time of testing for the control group
  years | 50 (12) | 45 (3) | 70 (7) | 58 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 2 | 11 | 25
  Male | 8 | 1 | 9 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 3 | 20 | 43
Duration of Hearing Loss [Mean (Standard Deviation); unit: years] | 3 (2) | 4 (2) | 3 (3) | 3 (2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Word Recognition in Quiet Over Time
Description: Results on recorded speech perception materials: monosyllabic (Consonant-Nucleus-Consonant) words in quiet during the first year of device use.
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: Three participants with asymmetric hearing loss did not complete the 9-month interval. One participant with asymmetric hearing loss withdrew from the study prior to the 12-month interval.
Measure: Mean (Standard Deviation); unit: percentage of words correctly repeated
Groups:
- Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group: Cochlear implantation of the affected ear
  Cochlear Implant: cochlear implantation used a treatment for unilateral hearing loss/single-sided deafness and/or asymmetric hearing loss
- Cochlear Implant: Asymmetric Hearing Loss Group: Cochlear implantation of the poorer hearing ear
  Cochlear Implant: cochlear implantation used a treatment for unilateral hearing loss/single-sided deafness and/or asymmetric hearing loss
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
percentage of words correctly repeated
  Before surgery, unaided | 4 (7) | 8 (11)
  1 month after surgery, unaided | 0 (1) | 0 (0)
  1 month after surgery, aided (cochlear implant) | 36 (18) | 32 (19)
  3 months after surgery, unaided | 0 (0) | 0 (0)
  3 months after surgery, aided (cochlear implant) | 47 (19) | 40 (17)
  6 months after surgery, unaided | 0 (1) | 0 (1)
  6 months after surgery, aided (cochlear implant) | 51 (15) | 47 (17)
  9 months after surgery, unaided: number analyzed (Participants) | 20 | 17
  9 months after surgery, unaided | 0 (0) | 0 (1)
  9 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 17
  9 months after surgery, aided (cochlear implant) | 55 (19) | 49 (22)
  12 months after surgery, unaided: number analyzed (Participants) | 20 | 19
  12 months after surgery, unaided | 0 (0) | 0 (0)
  12 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 19
  12 months after surgery, aided (cochlear implant) | 55 (18) | 55 (18)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Recorded 50-word consonant-nucleus-consonant (CNC) words were evaluated for the poorer hearing ear 1) unaided and 2) with the cochlear implant (CI) over the post-activation study period. A repeated-measures ANOVA evaluated the main effects of interval (1, 3, 6, 9, and 12 months post-activation), condition (unaided or with the CI), and their interaction. Percent correct converted to RAU; Test type: Superiority; p < 0.001, Mixed Models Analysis — Percent correct converted to rationalized arcsine units (RAU) prior to analysis; Main effects: interval (p<0.001) and condition (p<0.001). Interaction: Interval and condition (p<0.001)
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; Recorded 50-word CNC words were evaluated for the poorer hearing ear 1) unaided and 2) with the cochlear implant (CI) over the post-activation study period. A repeated-measures ANOVA evaluated the main effects of interval (1, 3, 6, 9, and 12 months post-activation), condition (unaided or with the CI), and their interaction. Percent correct converted to RAU; Test type: Superiority; p < 0.001, Mixed Models Analysis — Percent correct converted to rationalized arcsine units (RAU) prior to analysis; Main effects: interval (p<0.001) and condition (p<0.001). Interaction: interval and condition (p<0.001)
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Recorded 50-word CNC words were evaluated in an unaided condition for the poorer hearing ear pre-operatively and with the cochlear implant (CI) over the study period. A repeated-measures ANOVA evaluated the main effect of interval (before surgery, and 1, 3, 6, 9, and 12 months post-activation). Percent correct converted to RAU; Test type: Superiority; p < 0.001, ANOVA — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis; A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < 0.001, ANOVA — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis
Statistical Analysis 5: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group vs Cochlear Implant: Asymmetric Hearing Loss Group; Comparison of word recognition between groups (UHL/SSD and AHL) over the post-activation intervals (1, 3, 6, 9, and 12 months); Test type: Superiority; p < 0.429, Mixed Models Analysis — A logit transformation was applied to proportion correct data prior to analysis; Main effects: interval (p<0.001) and group (p=0.429). Interaction: group and interval (p=0.387)

2. Primary Outcome: Change in Localization Results (Measured in Root-mean-squared (RMS) Error) Over Time
Description: Subjects were asked to identify the noise source from an 11-speaker array with the cochlear implant on versus off. The intensity level of the stimulus was randomly varied (10 dB around 70 dB SPL) to limit the listener relying on level effects. Responses at each intensity level (i.e., 60, 70, and 80 dB SPL) for a given sound source (speaker) were combined (averaged). Results are reported in root-mean-squared (RMS) error. A lower value indicates better performance. Results are compared during the first year of cochlear implant use.
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: Three participants in the asymmetric hearing loss group did not complete the 9-month interval. One participant in the asymmetric hearing loss group withdrew from the study prior to the 12-month interval.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
degrees
  Before surgery, unaided | 67 (19) | 76 (19)
  1 month after surgery, unaided | 70 (19) | 79 (14)
  1 month after surgery, aided (cochlear implant) | 37 (19) | 52 (13)
  3 months after surgery, unaided | 68 (18) | 77 (15)
  3 months after surgery, aided (cochlear implant) | 28 (8) | 48 (10)
  6 months after surgery, unaided | 68 (18) | 79 (15)
  6 months after surgery, aided (cochlear implant) | 27 (7) | 43 (9)
  9 months after surgery, unaided: number analyzed (Participants) | 20 | 17
  9 months after surgery, unaided | 69 (19) | 78 (16)
  9 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 17
  9 months after surgery, aided (cochlear implant) | 26 (6) | 41 (9)
  12 months after surgery, unaided: number analyzed (Participants) | 20 | 19
  12 months after surgery, unaided | 67 (18) | 79 (17)
  12 months after surgery, aided (cochlear implant) | 27 (6) | 40 (11)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 60, 70, or 80 decibel (dB) sound pressure level (SPL) in a sound treated room. Overall root-mean-square (RMS) error is the difference between the sound source azimuth and the response azimuth and a lower score indicates more accurate localization of the sound source. A repeated-measures ANOVA evaluated the effects of interval, condition (unaided or with the cochlear implant), and their interaction; Test type: Superiority; p < 0.019, Mixed Models Analysis — The Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Main effects: interval (p=0.19) and condition (p<0.001). Interaction: interval and condition (p<0.019)
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.012, Mixed Models Analysis — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Main effects: interval (p=0.012) and condition (p<0.001). Interaction: interval and condition (p=0.004)
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 60, 70, or 80 decibel (dB) sound pressure level (SPL) in a sound treated room. Overall root-mean-square (RMS) error is the difference between the sound source azimuth and the response azimuth and a lower score indicates more accurate localization of the sound source. A repeated-measures ANOVA evaluated the effect of interval (pre-operatively, 1, 3, 6, 9, and 12 months post). Pre-op: unaided, Post: bilateral; Test type: Superiority; p < 0.001, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 60, 70, or 80 decibel (dB) sound pressure level (SPL) in a sound treated room. Overall root-mean-square (RMS) error is the difference between the sound source azimuth and the response azimuth and a lower score indicates more accurate localization of the sound source. A repeated-measures ANOVA evaluated the effects of interval (pre-operatively, 1, 3, 6, 9, and 12 months post). Pre-op: unaided, Post: bilateral; Test type: Superiority; p < 0.001, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 5: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Association of age at implantation and sound source localization (RMS) at the 12-month interval with the cochlear implant, analyzed with a Bivariate Pearson correlation (one-tailed); Test type: Other — correlation; p = 0.033, bivariate pearson correlation; bivariate pearson correlation = 0.42
Statistical Analysis 6: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group vs Cochlear Implant: Asymmetric Hearing Loss Group; Comparison of sound source localization between groups (UHL/SSD and AHL) over the post-activation intervals (1, 3, 6, 9, and 12 months); Test type: Superiority; p < 0.249, Mixed Models Analysis — There were significant main effects of group (p<0.001) and interval (p<0.001). There was a non-significant interaction between group and interval (p=0.249); Main effects: group (p<0.001) and interval (p<0.001). Interaction: group and interval (p=0.249)

3. Primary Outcome: Change in Subjective Benefit (Measured With the Speech, Spatial, and Qualities (SSQ) of Hearing Questionnaire) Over Time
Description: Subjects completed subjective questionnaires in order to evaluate the perceived benefits of cochlear implantation. For the Speech, Spatial, and Qualities of hearing questionnaire, participants rank their perceived abilities on a scale of 0-10. Higher values indicate more perceived abilities. Results are reported as the total score at each interval, which is the average of the responses from all questions for the questionnaire.
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: Three participants in the asymmetric hearing loss group did not complete the 9 month interval. One participant in the asymmetric hearing loss group withdrew from the study prior to the 12-month interval.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
score on a scale
  before surgery | 4 (1) | 4 (1)
  1 month after surgery | 6 (2) | 5 (1)
  3 months after surgery | 6 (2) | 6 (2)
  6 months after surgery | 7 (1) | 6 (1)
  9 months after surgery: number analyzed (Participants) | 20 | 17
  9 months after surgery | 7 (1) | 6 (1)
  12 months after surgery: number analyzed (Participants) | 20 | 19
  12 months after surgery | 7 (1) | 6 (1)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Responses on the Speech, Spatial, & Qualities of hearing scale (SSQ) as measured with the total score were compared over the post-activation period (i.e., 1, 3, 6, 9, and 12 months); Test type: Superiority; p < 0.001, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; Responses on the SSQ as measured with the total score were compared over the post-activation period (i.e., 1, 3, 6, 9, and 12 months); Test type: Superiority; p = 0.056, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Responses on the SSQ over the post-activation period (i.e., 1, 3, 6, 9, and 12 months). Subscales include: speech, spatial, and qualities of hearing. A repeated-measures ANOVA compared the main effects of interval and subscale and their interaction over time with the cochlear implant (1, 3, 6, 9, and 12 months post-activation); Test type: Superiority; p < 0.448, Mixed Models Analysis — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Main effects: interval (p<0.001) and subscale (p<0.001). Interaction: interval and subscale (p=0.488)
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.299, Mixed Models Analysis — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Main effects: subscale (p<0.001) and interval (p=0.072). Interaction: subscale and interval (p=0.299)
Statistical Analysis 5: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Responses on the SSQ Speech pragmatic subscale over the post-activation period (i.e., 1, 3, 6, 9, and 12 months). A repeated-measures ANOVA compared the main effects of interval and pragmatic subscale and their interaction over time with the cochlear implant (1, 3, 6, 9, and 12 months post-activation); Test type: Superiority; p < 0.018, Mixed Models Analysis — There were significant main effects of interval (p<0.001) and pragmatic subscale (p<0.001), and their interaction (p<0.018); Main effects: interval (p<0.001) and pragmatic subscale (p<0.001). Interaction: interval and pragmatic subscale (p<0.018)
Statistical Analysis 6: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Responses on the SSQ Spatial pragmatic subscale over the post-activation period (i.e., 1, 3, 6, 9, and 12 months). A repeated-measures ANOVA compared the main effects of interval and pragmatic subscale and their interaction over time with the cochlear implant (1, 3, 6, 9, and 12 months post-activation); Test type: Superiority; p < 0.767, Mixed Models Analysis; Main effects: interval (p<0.001) and pragmatic subscale (p=0.767). Interaction: interval and pragmatic subscale (p=0.542)
Statistical Analysis 7: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Responses on the SSQ Qualities of Hearing pragmatic subscale over the post-activation period (i.e., 1, 3, 6, 9, and 12 months). A repeated-measures ANOVA compared the main effects of interval and pragmatic subscale and their interaction over time with the cochlear implant (1, 3, 6, 9, and 12 months post-activation); Test type: Superiority; p < 0.242, Mixed Models Analysis; Main effects: interval (p=0.003) and pragmatic subscale (p<0.001). Interaction: interval and pragmatic subscale (p=0.242)
Statistical Analysis 8: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Association of subjective benefit (Speech Subscale) at the preoperative interval and speech recognition with AzBio sentences when the target is from the front and the masker is towards the acoustic ear; Test type: Other — Bivariate pearson correlation; p = 0.370, bivariate pearson correlation
Statistical Analysis 9: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 3, analysis 8]; Test type: Other — bivariate pearson correlation; p = 0.865, bivariate pearson correlation — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis
Statistical Analysis 10: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Association of subjective benefit (Speech Subscale) at the 12-month interval and speech recognition with AzBio sentences when the target is from the front and the masker is towards the acoustic ear; Test type: Other — bivariate pearson correlation; p = 0.005, bivariate pearson correlation — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis; bivariate pearson correlation = 0.60
Statistical Analysis 11: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 3, analysis 10]; Test type: Other — bivariate pearson correlation; p = 0.006, bivariate pearson correlation — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis; bivariate pearson correlation = 0.67
Statistical Analysis 12: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Association of subjective benefit (Spatial Subscale) at the preoperative interval and sound source localization (RMS error); Test type: Other — bivariate pearson correlation; p = 0.152, bivariate pearson correlation; bivariate pearson correlation = -0.33
Statistical Analysis 13: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 3, analysis 12]; Test type: Other — bivariate pearson correlation; p = 0.761, bivariate pearson correlation
Statistical Analysis 14: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Association of subjective benefit (Spatial Subscale) at the 12-month interval and sound source localization (RMS error); Test type: Other — bivariate pearson correlation; p = 0.315, bivariate pearson correlation
Statistical Analysis 15: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; Association of subjective benefit (Spatial Subscale) at the 12-month interval and sound source localization (RMS error); Test type: Other — bivariate pearson correlation; p = 0.666, bivariate pearson correlation
Statistical Analysis 16: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group vs Cochlear Implant: Asymmetric Hearing Loss Group; Comparison of subjective benefit between groups (UHL/SSD and AHL) on the speech, spatial, and qualities of hearing subscales during the post-activation intervals (1, 3, 6, 9, and 12 months); Test type: Superiority; p > 0.175, Mixed Models Analysis; Main effects: cohort (p=0.912), interval (p=0.463), and subscale (p=0.483). Interactions: 2-way or 3-way (p>0.175)

4. Primary Outcome: Change in Sentence Recognition in Noise Over Time, Measured With the AzBio Sentences With Speech Presented From the Front and Noise Towards the Better Hearing Ear
Description: Results on recorded speech perception materials: sentence recognition in noise with the target (speaker) from the front and the 10-talker masker 90 degrees towards the normal/better hearing ear. Scored as the percent correctly repeated.
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: Three participants with asymmetric hearing loss did not complete the 9-month interval. One participant with asymmetric hearing loss withdrew from the study prior to the 12-month interval. Four participants were tested at a different signal-to-noise ratio.
Measure: Mean (Standard Deviation); unit: percentage of words correctly repeated
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
percentage of words correctly repeated
  Before surgery, unaided: number analyzed (Participants) | 20 | 13
  Before surgery, unaided | 16 (13) | 3 (3)
  1 month after surgery, unaided: number analyzed (Participants) | 20 | 16
  1 month after surgery, unaided | 21 (14) | 5 (5)
  1 month after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 16
  1 month after surgery, aided (cochlear implant) | 40 (16) | 8 (8)
  3 months after surgery, unaided: number analyzed (Participants) | 20 | 16
  3 months after surgery, unaided | 25 (16) | 3 (6)
  3 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 16
  3 months after surgery, aided (cochlear implant) | 49 (19) | 10 (10)
  6 months after surgery, unaided: number analyzed (Participants) | 20 | 16
  6 months after surgery, unaided | 23 (18) | 2 (4)
  6 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 16
  6 months after surgery, aided (cochlear implant) | 49 (16) | 15 (10)
  9 months after surgery, unaided: number analyzed (Participants) | 20 | 14
  9 months after surgery, unaided | 25 (17) | 2 (4)
  9 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 14
  9 months after surgery, aided (cochlear implant) | 52 (18) | 15 (12)
  12 months after surgery, unaided: number analyzed (Participants) | 20 | 19
  12 months after surgery, unaided | 21 (19) | 4 (8)
  12 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 19
  12 months after surgery, aided (cochlear implant) | 53 (21) | 22 (18)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Recorded AzBio sentences in a 10-talker masker were evaluated in 2 conditions: 1) unaided and 2) with the cochlear implant (CI) over the post-activation study period. A repeated-measures ANOVA evaluated the main effects of interval (1, 3, 6, 9, and 12 months post-activation), condition (unaided or with the CI), and their interaction; Test type: Superiority; p < 0.161, Mixed Models Analysis — Significant effect of interval (p=0.046) and of condition (p<0.001) and a non-significant interaction (p=0.161). Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis; Main effects: interval (p=0.046) and condition (p<0.001). Interaction: interval and condition (p=0.161)
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p > 0.107, Mixed Models Analysis — Significant effect of condition (p<0.001) and the interaction (p<0.001). Non-significant effect of interval (p=0.107). Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis; Main effects: condition (p<0.001) and interval p=0.107). Interaction of condition and interval (p<0.001)
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Recorded AzBio sentences in a 10-talker masker were evaluated in an unaided condition for the poorer hearing ear pre-operatively and with the cochlear implant (CI) over the study period. A repeated-measures ANOVA evaluated the main effect of interval (before surgery, and 1, 3, 6, 9, and 12 months post-activation). Percent correct converted to RAU; Test type: Superiority; p < 0.001, ANOVA — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p < 0.001, ANOVA — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis
Statistical Analysis 5: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Association of age at implantation and speech recognition in noise at the 12-month interval with the cochlear implant, analyzed with a Bivariate Pearson correlation; Test type: Other — bivariate pearson correlation; p = 0.580, bivariate pearson correlation — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis
Statistical Analysis 6: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group vs Cochlear Implant: Asymmetric Hearing Loss Group; Comparison of speech recognition between groups (UHL/SSD and AHL) for the three masker configurations (noise towards the better hearing ear, noise towards the poorer hearing ear, and noise from the front) and signal-to-noise ratio (SNR; 0, 5, or 10 dB SNR) over the post-activation intervals (1, 3, 6, 9, and 12 months); Test type: Superiority; p < 0.743, Mixed Models Analysis — A logit transformation was applied to proportion correct data prior to analysis; Effects: SNR (p=0.026) & masker condition (p<0.001). Interactions: cohort & condition (p<0.001), interval & condition (p=0.015). Others (p>0.140)
Statistical Analysis 7: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Association of word recognition and speech recognition in noise, analyzed with a Bivariate Pearson correlation. Scores were averaged between 3 and 12 months post-activation as an estimate of asymptotic performance; Test type: Other — pearson correlation; p = 0.036, bivariate pearson correlation — Percent correct converted to rationalized arcsine units (RAU) prior to analysis

5. Primary Outcome: Change in Localization Results (Measured in Variable Error) Over Time
Description: Subjects were asked to identify the noise source from an 11-speaker array with the cochlear implant on versus off. The intensity level of the stimulus was randomly varied (10 dB around 70 dB SPL) to limit the listener relying on level effects. Responses at each intensity level (i.e., 60, 70, and 80 dB SPL) for a given sound source (speaker) were combined (averaged). Results are reported in variable error. A lower value indicates better performance. Results are compared during the first year of cochlear implant use.
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
degrees
  Before surgery, unaided | 24 (16) | 29 (18)
  1 month after surgery, unaided | 26 (18) | 25 (14)
  1 month after surgery, aided (cochlear implant) | 23 (10) | 35 (13)
  3 months after surgery, unaided | 28 (16) | 23 (12)
  3 months after surgery, aided (cochlear implant) | 19 (7) | 33 (12)
  6 months after surgery, unaided | 23 (14) | 23 (13)
  6 months after surgery, aided (cochlear implant) | 19 (7) | 28 (9)
  9 months after surgery, unaided: number analyzed (Participants) | 20 | 17
  9 months after surgery, unaided | 25 (14) | 23 (14)
  9 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 17
  9 months after surgery, aided (cochlear implant) | 18 (7) | 29 (11)
  12 months after surgery, unaided: number analyzed (Participants) | 20 | 19
  12 months after surgery, unaided | 28 (15) | 24 (17)
  12 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 19
  12 months after surgery, aided (cochlear implant) | 18 (7) | 27 (10)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 60, 70, or 80 decibel (dB) sound pressure level (SPL) in a sound treated room. Variable error is the average of the standard deviation of the responses for each source and a lower score reflects a more consistently accurate response. A repeated-measures ANOVA evaluated the effects of interval, condition (unaided or with the cochlear implant), and their interaction; Test type: Superiority; p < 0.183, Mixed Models Analysis — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Main effect: interval (p=0.183) and condition (p=0.012). Interaction: interval and condition (p=0.081)
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.196, Mixed Models Analysis — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Main effect: interval (p=0.010) and condition (p=0.100). Interaction: interval and condition (p=0.196)
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 60, 70, or 80 decibel (dB) sound pressure level (SPL) in a sound treated room. Variable error is the average of the standard deviation of the responses for each source and a lower score reflects a more consistently accurate response. A repeated-measures ANOVA evaluated the effect of interval (pre-operatively, 1, 3, 6, 9, and 12 months post). Pre-op: unaided, Post: bilateral; Test type: Superiority; p = 0.056, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 60, 70, or 80 decibel (dB) sound pressure level (SPL) in a sound treated room. Variable error is the average of the standard deviation of the responses for each source and a lower score reflects a more consistently accurate response. A repeated-measures ANOVA evaluated the effects of interval (pre-operatively, 1, 3, 6, 9, and 12 months post). Pre-op: unaided, Post: bilateral; Test type: Superiority; p = 0.210, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity

6. Primary Outcome: Change in Localization Results (Measured in Constant Error) Over Time
Description: Subjects were asked to identify the noise source from an 11-speaker array with the cochlear implant on versus off. The intensity level of the stimulus was randomly varied (10 dB around 70 dB SPL) to limit the listener relying on level effects. Responses at each intensity level (i.e., 60, 70, and 80 dB SPL) for a given sound source (speaker) were combined (averaged). Results are reported in constant error. A lower value indicates better performance. Results are compared during the first year of cochlear implant use.
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
degrees
  Before surgery, unaided | 59 (23) | 67 (24)
  1 month after surgery, unaided | 60 (24) | 73 (19)
  1 month after surgery, aided (cochlear implant) | 29 (18) | 37 (12)
  3 months after surgery, unaided | 58 (21) | 71 (18)
  3 months after surgery, aided (cochlear implant) | 20 (6) | 33 (9)
  6 months after surgery, unaided | 60 (23) | 74 (19)
  6 months after surgery, aided (cochlear implant) | 19 (7) | 31 (8)
  9 months after surgery, unaided: number analyzed (Participants) | 20 | 17
  9 months after surgery, unaided | 62 (23) | 72 (20)
  9 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 17
  9 months after surgery, aided (cochlear implant) | 18 (5) | 29 (7)
  12 months after surgery, unaided: number analyzed (Participants) | 20 | 19
  12 months after surgery, unaided | 58 (22) | 73 (21)
  12 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 19
  12 months after surgery, aided (cochlear implant) | 19 (5) | 28 (8)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 60, 70, or 80 decibel (dB) sound pressure level (SPL) in a sound treated room. Constant error is a measure of side bias, and a lower score indicates less response bias to either side. A repeated-measures ANOVA evaluated the effects of interval, condition (unaided or with the cochlear implant), and their interaction; Test type: Superiority; p < 0.071, Mixed Models Analysis — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Main effects: interval (p<0.071) and condition (p<0.001). Interaction: interval and condition (p<0.051)
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.109, Mixed Models Analysis — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Main effects: interval (p=0.109) and condition (p<0.001). Interaction: interval and condition (p=0.052)
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 60, 70, or 80 decibel (dB) sound pressure level (SPL) in a sound treated room. Constant error is a measure of side bias, and a lower score indicates less response bias to either side. A repeated-measures ANOVA evaluated the effect of interval (pre-operatively, 1, 3, 6, 9, and 12 months post). Pre-op: unaided, Post: bilateral; Test type: Superiority; p < 0.001, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 60, 70, or 80 decibel (dB) sound pressure level (SPL) in a sound treated room. Constant error is a measure of side bias, and a lower score indicates less response bias to either side. A repeated-measures ANOVA evaluated the effects of interval (pre-operatively, 1, 3, 6, 9, and 12 months post). Pre-op: unaided, Post: bilateral; Test type: Superiority; p < 0.001, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity

7. Primary Outcome: Change in Localization Results (Measured in Adjusted Constant Error) Over Time
Description: Subjects were asked to identify the noise source from an 11-speaker array with the cochlear implant on versus off. The intensity level of the stimulus was randomly varied (10 dB around 70 dB SPL) to limit the listener relying on level effects. Responses at each intensity level (i.e., 60, 70, and 80 dB SPL) for a given sound source (speaker) were combined (averaged). Results are reported in adjusted constant error. A lower value indicates better performance. Results are compared during the first year of cochlear implant use.
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
degrees
  Before surgery, unaided | 48 (9) | 48 (10)
  1 month after surgery, unaided | 47 (11) | 53 (6)
  1 month after surgery, aided (cochlear implant) | 23 (10) | 30 (8)
  3 months after surgery, unaided | 46 (12) | 52 (5)
  3 months after surgery, aided (cochlear implant) | 18 (5) | 29 (6)
  6 months after surgery, unaided | 47 (12) | 52 (5)
  6 months after surgery, aided (cochlear implant) | 16 (5) | 27 (7)
  9 months after surgery, unaided: number analyzed (Participants) | 20 | 17
  9 months after surgery, unaided | 47 (12) | 53 (5)
  9 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 17
  9 months after surgery, aided (cochlear implant) | 16 (5) | 26 (6)
  12 months after surgery, unaided: number analyzed (Participants) | 20 | 19
  12 months after surgery, unaided | 46 (12) | 53 (4)
  12 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 19
  12 months after surgery, aided (cochlear implant) | 16 (5) | 25 (6)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 60, 70, or 80 decibel (dB) sound pressure level (SPL) in a sound treated room. Adjusted constant error is a measure of reliability in the response taking side bias into account, and a lower score indicates a more reliable response. A repeated-measures ANOVA evaluated the effects of interval, condition (unaided or with the cochlear implant), and their interaction; Test type: Superiority; p < 0.024, Mixed Models Analysis — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Main effects: interval (p=0.018) and condition (p<0.001). Interaction: interval and condition (p=0.024)
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.219, Mixed Models Analysis; Main effects: interval (p=0.187) and condition (p<0.001). Interaction: interval and condition (p=0.219)
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 60, 70, or 80 decibel (dB) sound pressure level (SPL) in a sound treated room. Adjusted constant error is a measure of reliability in the response taking side bias into account, and a lower score indicates a more reliable response. A repeated-measures ANOVA evaluated the effect of interval (pre-operatively, 1, 3, 6, 9, and 12 months post). Pre-op: unaided, Post: bilateral; Test type: Superiority; p < 0.001, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 60, 70, or 80 decibel (dB) sound pressure level (SPL) in a sound treated room. Adjusted constant error is a measure of reliability in the response taking side bias into account, and a lower score indicates a more reliable response. A repeated-measures ANOVA evaluated the effects of interval (pre-operatively, 1, 3, 6, 9, and 12 months post). Pre-op: unaided, Post: bilateral; Test type: Superiority; p < 0.001, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity

8. Primary Outcome: Change in Subjective Benefit (Measured With the Abbreviated Profile of Hearing Aid Benefit (APHAB) Questionnaire) Over Time
Description: Subjects completed subjective questionnaires in order to evaluate the perceived benefits of cochlear implantation. For the Abbreviated Profile of Hearing Aid Benefit, participants rank their perceived difficulty on a scale of 1-99, with lower values indicate less perceived difficulty. The global score is average response across questions for the ease of communication, reverberation, and effectiveness in background noise subscales.
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
score on a scale
  before surgery | 50 (19) | 52 (17)
  1 month after surgery | 26 (13) | 32 (10)
  3 months after surgery | 21 (9) | 28 (10)
  6 months after surgery | 20 (8) | 31 (14)
  9 months after surgery: number analyzed (Participants) | 20 | 17
  9 months after surgery | 17 (8) | 29 (15)
  12 months after surgery: number analyzed (Participants) | 20 | 19
  12 months after surgery | 18 (9) | 28 (10)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Responses on the Abbreviated Profile of Hearing Aid Benefit (APHAB) as measured with the global score were compared over the post-activation period (i.e., 1, 3, 6, 9, and 12 months); Test type: Superiority; p = 0.011, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; The Abbreviated Profile of Hearing Aid Benefit, participants rank their perceived difficulty on a scale of 1-99, with lower values indicate less perceived difficulty. The global score is calculated from the responses on the ease of communication, reverberation, and effectiveness in background noise subscales. Responses were compared to responses over the post-activation period (1, 3, 6, 9, and 12 months) with the cochlear implant using a repeated-measures ANOVA; Test type: Superiority; p = 0.264, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; The Abbreviated Profile of Hearing Aid Benefit, participants rank their perceived difficulty on a scale of 1-99, with lower values indicate less perceived difficulty. Subscales include: ease of communication, reverberation, effectiveness in background noise, and reverberation. A repeated-measures ANOVA compared the main effects of interval and subscale and their interaction over time with the cochlear implant (1, 3, 6, 9, and 12 months post-activation); Test type: Superiority; p < 0.023, Mixed Models Analysis — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Main effects: interval (p=0.005) and subscales (p=0.001). Interaction: interval and subscales (p=0.023)
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p < 0.643, Mixed Models Analysis; Main effects: interval (p=0.643) and subscale (p=0.005). Interaction: interval and subscale (p=0.480)
Statistical Analysis 5: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Association of subjective benefit (Noise Subscale) at the preoperative interval and speech recognition with AzBio sentences when the target is from the front and the masker is towards the acoustic ear; Test type: Other — bivariate pearson correlation (one-tailed); p = 0.947, bivariate pearson correlation — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis
Statistical Analysis 6: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.500, bivariate pearson correlation — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis
Statistical Analysis 7: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Association of subjective benefit (Noise Subscale) at the 12-month interval and speech recognition with AzBio sentences when the target is from the front and the masker is towards the acoustic ear; Test type: Other — bivariate pearson correlation; p = 0.023, bivariate pearson correlation — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis; bivariate pearson correlation = -0.51
Statistical Analysis 8: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 8, analysis 7]; Test type: Other — bivariate pearson correlation; p = 0.033, bivariate pearson correlation — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis; bivariate pearson correlation = -0.55
Statistical Analysis 9: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group vs Cochlear Implant: Asymmetric Hearing Loss Group; Comparison of subjective benefit between groups (UHL/SSD and AHL) on the ease of communication, background noise, and reverberation subscales over the post-activation intervals (1, 3, 6, 9, and 12 months); Test type: Superiority; p > 0.208, Mixed Models Analysis; Main effects: cohort (p=0.541), interval (p=0.446), and subscale (p=0.208). Interactions: 2-way or 3-way (p>0.287)

9. Primary Outcome: Change in Subjective Benefit (Measured With the Tinnitus Handicap Inventory (THI) of Hearing Questionnaire) Over Time
Description: Subjects completed subjective questionnaires to order to evaluate the perceived benefits of cochlear implantation. For the Tinnitus Handicap Inventory, participants rank their perceived tinnitus severity on a scale of 0-100, with lower values indicate less tinnitus severity. Responses across all questions are summed to derive the total score.
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
score on a scale
  before surgery | 25 (17) | 18 (20)
  1 month after surgery | 6 (10) | 4 (6)
  3 months after surgery | 4 (7) | 2 (7)
  6 months after surgery | 2 (5) | 4 (12)
  9 months after surgery: number analyzed (Participants) | 20 | 17
  9 months after surgery | 4 (6) | 2 (7)
  12 months after surgery: number analyzed (Participants) | 20 | 19
  12 months after surgery | 3 (5) | 4 (13)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; The Tinnitus Handicap Inventory is a 25-item questionnaire. The subject answers "yes" (4 points), "sometimes" (2 points), or "no" (0 points) to each question. Responses are added to quantify tinnitus severity: none/slight (0-16), mild (18-36), moderate (38-56), severe (58-76), and catastrophic (78-100). Responses were compared over the post-activation time period (1, 3, 6, 9, and 12 months); Test type: Superiority; p = 0.221, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.538, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group vs Cochlear Implant: Asymmetric Hearing Loss Group; Comparison of subjective benefit between groups (UHL/SSD and AHL) on the Tinnitus Handicap Inventory over the post-activation intervals (1, 3, 6, 9, and 12 months); Test type: Superiority; p > 0.218, Mixed Models Analysis — There were no significant main effects of cohort (p=0.265) or interval (p=0.430). There was no significant interaction between cohort and interval (p=0.218); Main effects: cohort (p=0.265) or interval (p=0.430). Interaction: cohort and interval (p=0.218)

10. Primary Outcome: Change in Sentence Recognition in Noise Over Time, Measured With AzBio Sentences With Speech Presented From the Front and Noise Towards the Poorer Hearing Ear (Implanted Ear)
Description: Results on recorded speech perception materials: sentence recognition in noise with the target (speaker) from the front and the 10-talker masker 90 degrees towards the poorer hearing ear (implanted ear). Scored as the percent correctly repeated.
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of words correctly repeated
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
percentage of words correctly repeated
  Before surgery, unaided: number analyzed (Participants) | 20 | 13
  Before surgery, unaided | 83 (10) | 40 (18)
  1 month after surgery, unaided: number analyzed (Participants) | 20 | 16
  1 month after surgery, unaided | 88 (9) | 53 (17)
  1 month after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 16
  1 month after surgery, aided (cochlear implant) | 87 (7) | 49 (15)
  3 months after surgery, unaided: number analyzed (Participants) | 20 | 16
  3 months after surgery, unaided | 85 (9) | 39 (16)
  3 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 16
  3 months after surgery, aided (cochlear implant) | 87 (8) | 41 (18)
  6 months after surgery, unaided: number analyzed (Participants) | 20 | 16
  6 months after surgery, unaided | 89 (9) | 29 (19)
  6 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 16
  6 months after surgery, aided (cochlear implant) | 88 (7) | 38 (22)
  9 months after surgery, unaided: number analyzed (Participants) | 20 | 14
  9 months after surgery, unaided | 84 (15) | 38 (17)
  9 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 14
  9 months after surgery, aided (cochlear implant) | 89 (9) | 42 (21)
  12 months after surgery, unaided: number analyzed (Participants) | 20 | 15
  12 months after surgery, unaided | 84 (11) | 38 (24)
  12 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 15
  12 months after surgery, aided (cochlear implant) | 85 (11) | 42 (22)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.322, Mixed Models Analysis — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis; Main effect: interval (p=0.084) and condition (p=0.322). Interaction: interval and condition (p=0.125)
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.317, Mixed Models Analysis — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis; Main effects: interval (p=0.014) and condition (p=0.317). Interaction: interval and condition (p=0.118)
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.017, ANOVA — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.292, ANOVA — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis
Statistical Analysis 5: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; [analysis description as in outcome 4, analysis 7]; Test type: Other — pearson correlation; p > 0.185, bivariate pearson correlation

11. Primary Outcome: Change in Sentence Recognition in Noise Over Time, Measured With AzBio Sentences With Speech and Noise Presented From the Front
Description: Results on recorded speech perception materials: sentence recognition in noise with the target (speaker) and the 10-talker masker from the front speaker. Scored as the percent correctly repeated.
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of words correctly repeated
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
percentage of words correctly repeated
  Before surgery, unaided: number analyzed (Participants) | 20 | 13
  Before surgery, unaided | 37 (11) | 18 (12)
  1 month after surgery, unaided: number analyzed (Participants) | 20 | 16
  1 month after surgery, unaided | 39 (8) | 23 (14)
  1 month after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 16
  1 month after surgery, aided (cochlear implant) | 41 (8) | 28 (14)
  3 months after surgery, unaided: number analyzed (Participants) | 20 | 16
  3 months after surgery, unaided | 43 (10) | 17 (10)
  3 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 16
  3 months after surgery, aided (cochlear implant) | 45 (15) | 23 (10)
  6 months after surgery, unaided: number analyzed (Participants) | 20 | 16
  6 months after surgery, unaided | 38 (13) | 21 (14)
  6 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 16
  6 months after surgery, aided (cochlear implant) | 45 (10) | 26 (10)
  9 months after surgery, unaided: number analyzed (Participants) | 20 | 14
  9 months after surgery, unaided | 45 (15) | 20 (15)
  9 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 14
  9 months after surgery, aided (cochlear implant) | 49 (12) | 25 (14)
  12 months after surgery, unaided: number analyzed (Participants) | 20 | 15
  12 months after surgery, unaided | 42 (12) | 22 (15)
  12 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 15
  12 months after surgery, aided (cochlear implant) | 47 (11) | 24 (14)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.581, Mixed Models Analysis — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis; Main effect: interval (p=0.039) and condition (p=0.007). Interaction: interval and condition (p=0.581)
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.817, Mixed Models Analysis — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis; Main effects: condition (p=0.005) and interval (p=0.528). Interaction: condition and interval (p=0.817)
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.008, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.009, ANOVA
Statistical Analysis 5: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Association of age at implantation and performance at the 12-month interval with the cochlear implant, analyzed with a Bivariate Pearson correlation (one-tailed); Test type: Other — bivariate correlation; p = 0.049, bivariate pearson correlation — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis. This correlation was no longer significant when controlling for the hearing threshold at 8000 Hz
Statistical Analysis 6: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; [analysis description as in outcome 4, analysis 7]; Test type: Other — pearson correlation; p > 0.185, bivariate pearson correlation

12. Primary Outcome: Change in Sentence Recognition in Noise Over Time, Measured With Bamford-Kowal-Bamford (BKB) Sentences With Speech and Noise Presented From the Front
Description: Results on recorded speech perception materials: sentence recognition in noise with the target (speaker) and the 4-talker masker from the front speaker. Scored as dB signal-to-noise ratio that the listener gets 50% speech understanding. Lower numbers indicate better performance (range -7.5 to 23.5 dB SNR).
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: signal-to-noise ratio
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
signal-to-noise ratio
  Before surgery, unaided | 0.2 (1.4) | 4.2 (3.5)
  1 month after surgery, unaided | -0.2 (1.2) | 3.3 (4.1)
  1 month after surgery, aided (cochlear implant) | -0.6 (1.5) | 2.6 (3.1)
  3 months after surgery, unaided | -0.2 (1.3) | 3.6 (3.8)
  3 months after surgery, aided (cochlear implant) | -0.9 (1.7) | 2.6 (3.1)
  6 months after surgery, unaided | -0.1 (2.4) | 3.1 (3.8)
  6 months after surgery, aided (cochlear implant) | -0.9 (1.4) | 1.8 (3.6)
  9 months after surgery, unaided: number analyzed (Participants) | 20 | 16
  9 months after surgery, unaided | -0.7 (1.4) | 2.7 (2.7)
  9 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 16
  9 months after surgery, aided (cochlear implant) | -1.4 (1.4) | 1.4 (2.5)
  12 months after surgery, unaided: number analyzed (Participants) | 20 | 19
  12 months after surgery, unaided | -0.9 (1.2) | 3.9 (3.7)
  12 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 19
  12 months after surgery, aided (cochlear implant) | -0.8 (1.7) | 3.4 (3.4)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Recorded BKB sentences in a 4-talker masker were evaluated in 2 conditions: 1) unaided and 2) with the cochlear implant (CI) over the post-activation study period. Results are reported in dB SNR, where a lower value indicates better performance. A repeated-measures ANOVA evaluated the main effects of interval (1, 3, 6, 9, and 12 months post-activation), condition (unaided or with the CI), and their interaction; Test type: Superiority; p < 0.440, Mixed Models Analysis; Main effects: interval (p=0.070) and condition (p=0.440). Interaction: interval and condition (p=0.047)
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.379, Mixed Models Analysis; Main effects: condition (p<0.001) and interval (p=0.250). Interaction: interval and condition (p=0.379)
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Recorded BKB sentences in a 4-talker masker were evaluated in an unaided condition for the poorer hearing ear pre-operatively and with the cochlear implant (CI) over the study period. A repeated-measures ANOVA evaluated the main effect of interval (before surgery, and 1, 3, 6, 9, and 12 months post-activation); Test type: Superiority; p = 0.021, ANOVA
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 12, analysis 3]; Test type: Superiority; p < 0.001, ANOVA

13. Primary Outcome: Change in Sentence Recognition in Noise Over Time, Measured With Bamford-Kowal-Bamford (BKB) Sentences With Speech Presented From the Front and Noise Towards the Better Hearing Ear
Description: Results on recorded speech perception materials: sentence recognition in noise with the target (speaker) from the front and the 4-talker masker 90 degrees towards the normal/better hearing ear. Scored as dB signal-to-noise ratio that the listener gets 50% speech understanding. A lower value indicates better performance (range -7.5 to 23.5 dB SNR).
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: signal-to-noise ratio
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
signal-to-noise ratio
  Before surgery, unaided | 1.8 (1.3) | 7.1 (4.0)
  1 month after surgery, unaided | 0.7 (1.8) | 6.8 (4.1)
  1 month after surgery, aided (cochlear implant) | -0.2 (2.2) | 5.2 (3.4)
  3 months after surgery, unaided | 0.6 (1.9) | 6.9 (3.5)
  3 months after surgery, aided (cochlear implant) | -1.0 (2.5) | 4.6 (3.3)
  6 months after surgery, unaided | 0.6 (1.7) | 6.9 (3.4)
  6 months after surgery, aided (cochlear implant) | -0.7 (1.1) | 3.9 (3.3)
  9 months after surgery, unaided: number analyzed (Participants) | 20 | 16
  9 months after surgery, unaided | 0.7 (2.0) | 6.2 (3.4)
  9 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 16
  9 months after surgery, aided (cochlear implant) | -1.2 (1.7) | 4.2 (3.0)
  12 months after surgery, unaided: number analyzed (Participants) | 20 | 19
  12 months after surgery, unaided | 0.8 (1.4) | 6.9 (4.2)
  12 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 19
  12 months after surgery, aided (cochlear implant) | -1.0 (2.2) | 4.4 (4.3)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.639, Mixed Models Analysis — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Main effect: condition (p<0.001) and interval (p=0.639). Interaction: interval and condition (p=0.280)
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.637, Mixed Models Analysis; Main effects: condition (p<0.001) and interval (p=0.637). Interaction: interval and condition (p=0.450)
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; [analysis description as in outcome 12, analysis 3]; Test type: Superiority; p < 0.001, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 12, analysis 3]; Test type: Superiority; p = 0.002, ANOVA

14. Primary Outcome: Change in Sentence Recognition in Noise Over Time, Measured With Bamford-Kowal-Bamford (BKB) Sentences With Speech Presented From the Front and Noise Towards the Poorer Hearing Ear (Implanted Ear)
Description: Results on recorded speech perception materials: sentence recognition in noise with the target (speaker) from the front and the 4-talker masker 90 degrees towards the poorer hearing ear (implanted ear). Scored as dB signal-to-noise ratio that the listener gets 50% speech understanding. Lower values indicate better performance (range -7.5 to 23.5 dB SNR).
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: signal-to-noise ratio
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
signal-to-noise ratio
  Before surgery, unaided | -4.8 (1.6) | 1.4 (3.8)
  1 month after surgery, unaided | -5.1 (1.0) | 0.4 (4.6)
  1 month after surgery, aided (cochlear implant) | -5.3 (1.5) | 0.5 (4.6)
  3 months after surgery, unaided | -5.2 (1.6) | 1.4 (4.2)
  3 months after surgery, aided (cochlear implant) | -5.0 (1.5) | 1.7 (3.6)
  6 months after surgery, unaided | -4.9 (1.3) | 1.4 (4.0)
  6 months after surgery, aided (cochlear implant) | -5.3 (1.5) | 1.3 (4.1)
  9 months after surgery, unaided: number analyzed (Participants) | 20 | 16
  9 months after surgery, unaided | -5.5 (1.2) | 0.5 (3.8)
  9 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 16
  9 months after surgery, aided (cochlear implant) | -5.9 (1.1) | 0.8 (3.6)
  12 months after surgery, unaided: number analyzed (Participants) | 20 | 19
  12 months after surgery, unaided | -4.7 (1.8) | 2.3 (4.9)
  12 months after surgery, aided (cochlear implant): number analyzed (Participants) | 20 | 19
  12 months after surgery, aided (cochlear implant) | -4.8 (1.7) | 2.4 (3.8)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.671, Mixed Models Analysis; Main effects: interval (p=0.020) and condition (p=0.406). Interaction: interval and condition (p=0.671)
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p > 0.124, Mixed Models Analysis; Main effects: interval (p=0.124) and condition (p=0.845). Interaction: interval and condition (p=0.960)
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; [analysis description as in outcome 12, analysis 3]; Test type: Superiority; p = 0.025, ANOVA
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 12, analysis 3]; Test type: Superiority; p = 0.442, ANOVA

15. Secondary Outcome: Aided Word Recognition With a Cochlear Implant Versus a Current Treatment Option (i.e., Hearing Aid)
Description: Results on recorded speech perception materials: aided word recognition. Recorded 50-word CNC words were evaluated preoperatively with a conventional hearing aid. Performance was compared to the CI alone at the 12 month interval. A paired samples t-test compared the performance with the two devices. Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis to control for potential floor or ceiling effects (e.g., scores <20%).
Time Frame: preoperative interval and 12 month post-activation interval
Population: One asymmetric hearing loss participant withdrew prior to the 12-month interval.
Measure: Mean (Standard Deviation); unit: percentage of words correct
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
percentage of words correct
  preop, hearing aid | 4 (7) | 8 (9)
  12-month post-activation, cochlear implant | 55 (18) | 55 (18)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Paired samples t-test comparing word recognition (percent correct for CNC words) with a hearing aid at the pre-operative interval and the cochlear implant at the 12-month interval for the affected ear (masking presented to the contralateral ear); Test type: Superiority; p < 0.001, t-test, 2 sided — Percent correct values were converted to rationalized arcsine units prior to analysis
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p < 0.001, t-test, 2 sided — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis

16. Secondary Outcome: Localization Abilities With a Cochlear Implant Versus a Current Treatment Option (i.e., Bone-conduction Device)
Description: Subjects were asked to identify the noise source from an 11-speaker array with the cochlear implant on versus with a bone-conduction device. The intensity level of the stimulus was randomly varied (10 dB around 70 dB SPL) to limit the listener relying on level effects. Responses at each intensity level (i.e., 60, 70, and 80 dB SPL) for a given sound source (speaker) were combined (averaged). Results are reported in root-mean-squared (RMS) error. A lower value indicates better performance.
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: Three participants in the asymmetric group did not complete testing at the 9-month interval. One participant did not complete testing with the CI on at the 12-month interval. Three participants did not complete testing in the with the bone conduction device at the 12-month interval.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
degrees
  preoperative, bone-conduction device | 70 (19) | 76 (18)
  1-month, cochlear implant | 37 (19) | 52 (13)
  3-month, cochlear implant | 28 (8) | 48 (10)
  6-month, cochlear implant | 27 (7) | 43 (9)
  9-month, cochlear implant: number analyzed (Participants) | 20 | 17
  9-month, cochlear implant | 26 (6) | 41 (9)
  12-month, cochlear implant: number analyzed (Participants) | 20 | 19
  12-month, cochlear implant | 27 (6) | 40 (11)
  12-month, bone conduction device: number analyzed (Participants) | 20 | 17
  12-month, bone conduction device | 69 (19) | 80 (14)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Participants listened with a bone conduction device preoperatively and with the cochlear implant at 1, 3, 6, 9, and 12 months post-activation. Overall root-mean-square (RMS) error is the difference between the sound source azimuth and the response azimuth and a lower score indicates more accurate localization of the sound source. Repeated-measures ANOVA compared performance over time; Test type: Superiority; p < 0.001, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; Participants listening with a bone conduction device preoperatively and with the cochlear implant at 1, 3, 6, 9, and 12 months post-activation. Overall root-mean-square (RMS) error is the difference between the sound source azimuth and the response azimuth and a lower score indicates more accurate localization of the sound source. Repeated-measures ANOVA compared performance over time; Test type: Superiority; p < 0.001, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Compare localization performance with the cochlear implant to a bone-conduction device at the 12-month interval using a paired samples t-test; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 16, analysis 3]; Test type: Superiority; p < 0.001, t-test, 2 sided

17. Secondary Outcome: Subjective Benefit (Measured With the Abbreviated Profile of Hearing Aid Benefit Questionnaire) With Cochlear Implant Versus Preoperative Perceptions With Alternative Treatment Options (e.g., Hearing Aid, Bone-conduction Device)
Description: Subjects completed subjective questionnaires. For the Abbreviated Profile of Hearing Aid Benefit, participants rank their perceived difficulty on a scale of 1-99, with lower values indicate less perceived difficulty. The global score is the average response across questions for the ease of communication, reverberation, and effectiveness in background noise subscales.
Time Frame: preoperative interval, and post-activation intervals (1, 3, 6, 9, and 12 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
score on a scale
  before surgery | 50 (19) | 52 (17)
  1 month after surgery | 26 (13) | 32 (10)
  3 months after surgery | 21 (9) | 28 (10)
  6 months after surgery | 20 (8) | 31 (14)
  9 months after surgery: number analyzed (Participants) | 20 | 17
  9 months after surgery | 17 (8) | 29 (15)
  12 months after surgery: number analyzed (Participants) | 20 | 19
  12 months after surgery | 18 (9) | 28 (10)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; The Abbreviated Profile of Hearing Aid Benefit, participants rank their perceived difficulty on a scale of 1-99, with lower values indicate less perceived difficulty. The global score is calculated from the responses on the ease of communication, reverberation, and effectiveness in background noise subscales. Responses at the preoperative interval (alternative treatments for unilateral hearing loss) were compared to responses over time with the cochlear implant using a repeated-measures ANOVA; Test type: Superiority; p < 0.001, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p < 0.001, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; The Abbreviated Profile of Hearing Aid Benefit, participants rank their perceived difficulty on a scale of 1-99, with lower values indicate less perceived difficulty. Subscales include: ease of communication, reverberation, effectiveness in background noise, and reverberation. A repeated-measures ANOVA compared the main effects of interval and subscale and their interaction from the preoperative interval (alternative treatments) and over time with the cochlear implant; Test type: Superiority; p < 0.001, Mixed Models Analysis — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Main effects: interval (p<0.001) and subscales (p<0.001). Interaction: interval and subscales (p<0.001)
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 17, analysis 3]; Test type: Superiority; p < 0.010, Mixed Models Analysis — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Main effects: interval (p<0.001) and subscales (p=0.010). Interaction: interval and subscales (p=0.001)

18. Secondary Outcome: Subjective Benefit (Measured With the Tinnitus Handicap Inventory (THI) Questionnaire) With Cochlear Implant Versus Preoperative Perceptions With Alternative Treatment Options (e.g., Hearing Aid, Bone-conduction Device)
Description: Subjects completed subjective questionnaires. For the Tinnitus Handicap Inventory, participants rank their perceived tinnitus severity on a scale of 0-100, with lower values indicate less tinnitus severity. Responses across all questions are summed to derive the total score.
Time Frame: Intervals within the first year of device use (e.g., preoperative, and 1-, 3-, 6-, 9-, and 12-months post-activation)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
score on a scale
  before surgery | 25 (17) | 18 (20)
  1 month after surgery | 6 (10) | 4 (6)
  3 months after surgery | 4 (7) | 2 (7)
  6 months after surgery | 2 (5) | 4 (12)
  9 months after surgery: number analyzed (Participants) | 20 | 17
  9 months after surgery | 4 (6) | 2 (7)
  12 months after surgery: number analyzed (Participants) | 20 | 19
  12 months after surgery | 3 (5) | 4 (13)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; The Tinnitus Handicap Inventory is a 25-item questionnaire. The subject answers "yes" (4 points), "sometimes" (2 points), or "no" (0 points) to each question. Responses are added to quantify tinnitus severity: none/slight (0-16), mild (18-36), moderate (38-56), severe (58-76), and catastrophic (78-100). Responses were compared at the preoperative interval (alternative treatments) and over the post-activation time period (1, 3, 6, 9, and 12 months) with the cochlear implant; Test type: Superiority; p < 0.001, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.003, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity

19. Secondary Outcome: Subjective Benefit (Measured With the Speech, Spatial, and Qualities of Hearing (SSQ) Questionnaire) With Cochlear Implant Versus Preoperative Perceptions With Alternative Treatment Options (e.g., Hearing Aid, Bone-conduction Device)
Description: Subjects completed subjective questionnaires. For the Speech, Spatial, and Qualities of hearing questionnaire, participants rank their perceived abilities on a scale of 0-10. Higher values indicate more perceived abilities. Results are reported as the total score at each interval, which is the average of the responses from all questions for the questionnaire.
Time Frame: preoperative interval, and post-activation intervals (1, 3, 6, 9, and 12 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
score on a scale
  before surgery | 4 (1) | 4 (1)
  1 month after surgery | 6 (2) | 5 (1)
  3 months after surgery | 6 (2) | 6 (2)
  6 months after surgery | 7 (1) | 6 (1)
  9 months after surgery: number analyzed (Participants) | 20 | 17
  9 months after surgery | 7 (1) | 6 (1)
  12 months after surgery: number analyzed (Participants) | 20 | 19
  12 months after surgery | 7 (1) | 6 (1)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Responses on the SSQ as measured with the total score were compared at the preoperative interval (alternative treatments for SSD) and over the post-activation period (i.e., 1, 3, 6, 9, and 12 months); Test type: Superiority; p < 0.001, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; Responses on the SSQ as measured with the total score were compared at the preoperative interval (alternative treatments for asymmetric hearing loss) and over the post-activation period (i.e., 1, 3, 6, 9, and 12 months); Test type: Superiority; p < 0.001, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity
Statistical Analysis 3: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Responses on the SSQ as measured with the subscales (speech, spatial, & qualities) were compared at the preoperative interval (alternative treatments for SSD) and over the post-activation period (i.e., 1, 3, 6, 9, and 12 months). A repeated-measures ANOVA assessed the main effects of interval and subscale, and their interaction; Test type: Superiority; p < 0.001, Mixed Models Analysis — There were significant main effects of interval (p<0.001) and subscale (p<0.001) and interaction (p=0.001). A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Main effects: interval (p<0.001) and subscale (p<0.001). Interaction: interval and subscale (p=0.001)
Statistical Analysis 4: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; Responses on the SSQ as measured with the subscales (speech, spatial, & qualities) were compared at the preoperative interval (alternative treatments for asymmetric hearing loss) and over the post-activation period (i.e., 1, 3, 6, 9, and 12 months). A repeated-measures ANOVA assessed the main effects of interval and subscale, and their interaction; Test type: Superiority; p < 0.034, Mixed Models Analysis — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Main effects: interval (p<0.001) and subscale (p<0.001). Interaction: interval and subscale (p=0.034)
Statistical Analysis 5: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Responses on the SSQ Speech pragmatic subscale over the study period (i.e., preoperative, and 1, 3, 6, 9, and 12 months post-activation). A repeated-measures ANOVA compared the main effects of interval and pragmatic subscale and their interaction over time; Test type: Superiority; p < 0.001, Mixed Models Analysis; Main effects: interval (p<0.001) and pragmatic subscale (p<0.001). Interaction: interval and pragmatic subscale (p<0.001)
Statistical Analysis 6: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Responses on the SSQ Spatial pragmatic subscale over the study period (i.e., preoperative, and 1, 3, 6, 9, and 12 months post-activation). A repeated-measures ANOVA compared the main effects of interval and pragmatic subscale and their interaction over time; Test type: Superiority; p < 0.192, Mixed Models Analysis; Main effect: interval (p<0.001) and pragmatic subscale (p=0.192). Interaction: interval and pragmatic subscale (p=0.001)
Statistical Analysis 7: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Responses on the SSQ Qualities of Hearing pragmatic subscale over the study period (i.e., preoperative, and 1, 3, 6, 9, and 12 months post-activation). A repeated-measures ANOVA compared the main effects of interval and pragmatic subscale and their interaction over time; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 19, analysis 5]
Statistical Analysis 8: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 19, analysis 5]; Test type: Superiority; p < 0.479, Mixed Models Analysis; Main effects: interval (p<0.001) and pragmatic subscale (p<0.001). Interaction: interval and pragmatic subscale (p=0.479)
Statistical Analysis 9: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 19, analysis 6]; Test type: Superiority; p < 0.804, Mixed Models Analysis; Main effect: interval (p<0.001) and pragmatic subscale (p=0.804). Interaction: interval and pragmatic subscale (p=0.090)
Statistical Analysis 10: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 19, analysis 7]; Test type: Superiority; p < 0.005, Mixed Models Analysis; Main effects: interval (p<0.001) and pragmatic subscale (p<0.001). Interaction: interval and pragmatic subscale (p=0.005)

20. Secondary Outcome: Speech Perception Outcomes With a Cochlear Implant Versus a Bone-conduction Device: Sentence Recognition in Noise (AzBio, Speech Front and Noise Front)
Description: Recorded AzBio sentences in a 10-talker masker were evaluated in 2 conditions: 1) bone-conduction device at the preoperative interval and 2) with the cochlear implant (CI) at the 12-month post-activation period. A paired samples t-test compared the performance with the two devices. Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis.
Time Frame: preoperative interval and 12 month post-activation interval
Population: One participant with asymmetric hearing loss withdrew from the study prior to the 12-month interval. Seven participants were tested at a different signal-to-noise ratio at the preoperative interval. Four participants were tested at a different signal-to-noise ratio.
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
percent correct
  pre-op, bone-conduction device: number analyzed (Participants) | 20 | 13
  pre-op, bone-conduction device | 32 (17) | 17 (12)
  12-month post-activation, cochlear implant: number analyzed (Participants) | 20 | 15
  12-month post-activation, cochlear implant | 47 (11) | 24 (14)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Recorded AzBio sentences in a 10-talker masker were evaluated in 2 conditions: 1) bone-conduction device at the preoperative interval and 2) with the cochlear implant (CI) at the 12-month post-activation period. A paired samples t-test compared the performance with the two devices. Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis; Test type: Superiority; p = 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.034, t-test, 2 sided

21. Secondary Outcome: Speech Perception Outcomes With a Cochlear Implant Versus a Bone-conduction Device: Sentence Recognition in Noise (AzBio, Speech Front and Noise to the Poorer Hearing Ear)
Description: as for outcome 20
Time Frame: preoperative interval and 12 month post-activation interval
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
percent correct
  pre-op, bone-conduction device: number analyzed (Participants) | 20 | 13
  pre-op, bone-conduction device | 61 (28) | 24 (18)
  12-month post-activation, cochlear implant | 85 (11) | 42 (22)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.037, t-test, 2 sided

22. Secondary Outcome: Speech Perception Outcomes With a Cochlear Implant Versus a Bone-conduction Device: Sentence Recognition in Noise (AzBio, Speech Front and Noise to the Better Hearing Ear)
Description: as for outcome 20
Time Frame: preoperative interval and 12 month post-activation interval
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
percent correct
  pre-op, bone-conduction device: number analyzed (Participants) | 20 | 13
  pre-op, bone-conduction device | 18 (18) | 6 (8)
  12-month post-activation, cochlear implant: number analyzed (Participants) | 20 | 15
  12-month post-activation, cochlear implant | 53 (21) | 22 (18)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.001, t-test, 2 sided

23. Secondary Outcome: Speech Perception Outcomes With a Cochlear Implant Versus a Bone-conduction Device: Sentence Recognition in Noise (BKB-Speech In Noise (SIN), Speech Front and Noise Front)
Description: Recorded BKB sentences in a 4-talker masker were evaluated in 2 conditions: 1) bone-conduction device at the preoperative interval and 2) with the cochlear implant (CI) at the 12-month post-activation period. A paired samples t-test compared the performance with the two devices. Results are reported in dB SNR, where a lower value indicates better performance (range -7.5 to 23.5 dB SNR).
Time Frame: preoperative interval and 12 month post-activation interval
Population: One asymmetric hearing loss participant withdrew prior to the 12-month interval.
Measure: Mean (Standard Deviation); unit: signal-to-noise ratio
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
signal-to-noise ratio
  pre-op, bone-conduction device | 0.8 (2.0) | 4.9 (3.0)
  12-month post-activation, cochlear implant: number analyzed (Participants) | 20 | 19
  12-month post-activation, cochlear implant | -0.8 (1.7) | 3.4 (3.4)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; Recorded BKB sentences in a 4-talker masker were evaluated in 2 conditions: 1) with a bone-conduction device (preoperative interval) and 2) with the cochlear implant (CI) at the 12-month post-activation interval. Results are reported in dB SNR, where a lower value indicates better performance. A paired samples t-test compared the performance with the two devices; Test type: Superiority; p = 0.004, t-test, 2 sided
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; Recorded BKB sentences in a 4-talker masker were evaluated in 2 conditions: 1) bone-conduction device at the preoperative interval and 2) with the cochlear implant (CI) at the 12-month post-activation period. A paired samples t-test compared the performance with the two devices. Results are reported in dB SNR, where a lower value indicates better performance; Test type: Superiority; p = 0.004, t-test, 2 sided

24. Secondary Outcome: Speech Perception Outcomes With a Cochlear Implant Versus a Bone-conduction Device: Sentence Recognition in Noise (BKB-SIN, Speech Front and Noise to the Poorer Hearing Ear)
Description: as for outcome 23
Time Frame: preoperative interval and 12 month post-activation interval
Population: One asymmetric hearing loss participant withdrew prior to the 12-month interval.
Measure: Mean (Standard Deviation); unit: signal-to-noise ratio
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
signal-to-noise ratio
  pre-op, bone-conduction device | -2.6 (2.4) | 2.7 (3.7)
  12-month post-activation, cochlear implant: number analyzed (Participants) | 20 | 19
  12-month post-activation, cochlear implant | -4.8 (1.7) | 2.4 (3.8)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; [analysis description as in outcome 23, analysis 2]; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 23, analysis 2]; Test type: Superiority; p = 0.727, t-test, 2 sided

25. Secondary Outcome: Speech Perception Outcomes With a Cochlear Implant Versus a Bone-conduction Device: Sentence Recognition in Noise (BKB-SIN, Speech Front and Noise to the Better Hearing Ear)
Description: as for outcome 23
Time Frame: preoperative interval and 12 month post-activation interval
Population: One asymmetric hearing loss participant withdrew prior to the 12-month interval.
Measure: Mean (Standard Deviation); unit: signal-to-noise ratio
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
signal-to-noise ratio
  pre-op, bone-conduction device | 1.8 (2.3) | 6.1 (4.4)
  12-month post-activation, cochlear implant: number analyzed (Participants) | 20 | 19
  12-month post-activation, cochlear implant | -1.0 (2.2) | 4.4 (4.3)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; [analysis description as in outcome 23, analysis 2]; Test type: Superiority; p = 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 23, analysis 2]; Test type: Superiority; p = 0.090, t-test, 2 sided

26. Secondary Outcome: Speech Recognition in Noise for a Control Group: AzBio Sentences (0 dB SNR)
Description: The speech perception (cochlear implant recipients with UHL/SSD) to a control group of implantable bone-conduction device recipients (alternative treatment option). Participants in the control group had at least 12 months of listening experience with their implanted bone-conduction device prior to study participation. Sentence recognition was assessed in a 10-talker masker at 0 dB SNR with the target speech presented from the front and the masker (1) presented from the front (SoNo), (2) presented towards the implanted ear (SoNbc), and (3) presented towards the acoustic ear (SoNnh). Performance was scored as the percent of words correctly repeated, with higher values indicating better performance. The task was completed with the participants listening with their bone-conduction device on versus off.
Time Frame: Assessment completed after 12 months of implantable bone-conduction listening experience
Population: Performance on measures of speech perception
Measure: Median (Full Range); unit: percentage of words correctly repeated
Groups:
- Control Group: Recipients of a Bone-conduction Device on the Affected Side: Recipients of an implantable bone-conduction device with at least 12 months of listening experience. Participants were adults (18 years of age or older) with a duration of moderate-to-profound hearing loss of 5 years or less at the time of implantation with a bone-conduction device and normal hearing to mild hearing loss in the contralateral ear.
Arm/Group | Control Group: Recipients of a Bone-conduction Device on the Affected Side
Number analyzed (Participants) | 3
percentage of words correctly repeated
  SoNo, device on | 32 [30 to 53]
  SoNbc, device on | 69 [68 to 72]
  SoNnh, device on | 10 [5 to 17]
  SoNo, device off | 19 [18 to 48]
  SoNbc, device off | 80 [69 to 89]
  SoNnh, device off | 7 [5 to 9]

27. Secondary Outcome: Speech Recognition in Noise for a Control Group: BKB-SIN Test
Description: The speech perception outcomes in the study population (cochlear implant recipients with UHL/SSD) to a control group of implantable bone-conduction device recipients (alternative treatment option). Participants in the control group had at least 12 months of listening experience with their implanted bone-conduction device prior to study participation. Sentence recognition was assessed in a 4-talker masker with the target speech presented from the front and the masker (1) presented from the front, (2) presented towards the implanted ear, and (3) presented towards the acoustic ear. Performance was scored as the dB SNR when the participant understood 50% correct, with lower values indicating better performance. Participants completed the task with the device on and off.
Time Frame: Assessment completed after 12 months of implantable bone-conduction listening experience
Measure: Median (Full Range); unit: signal-to-noise ratio
Arm/Group | Control Group: Recipients of a Bone-conduction Device on the Affected Side
Number analyzed (Participants) | 3
signal-to-noise ratio
  SoNo, device on | -1 [-1 to 0]
  SoNbc, device on | -2.5 [-4.5 to -2]
  SoNnh, device on | 2 [-1 to 2.5]
  SoNo, device off | -1 [-2 to 2]
  SoNbc, device off | -4.5 [-6 to -4]
  SoNnh, device off | 3 [1.5 to 4.5]

28. Secondary Outcome: Localization for a Control Group
Description: Subjects were asked to identify the noise source from an 11-speaker array with the bone-conduction device on versus off. The intensity level of the stimulus was randomly varied (10 dB around 70 dB SPL) to limit the listener relying on level effects. Responses at each intensity level (i.e., 60, 70, and 80 dB SPL) for a given sound source (speaker) were combined (averaged). Results are reported in root-mean-squared (RMS) error. A lower value indicates better performance. Subjects in the control group were implantable bone-conduction device recipients (alternative treatment option) with at least 12 months of listening experience with their implanted bone-conduction device. Participants completed the task with their device on and off.
Time Frame: Assessment completed after 12 months of implantable bone-conduction listening experience
Measure: Median (Full Range); unit: degrees
Arm/Group | Control Group: Recipients of a Bone-conduction Device on the Affected Side
Number analyzed (Participants) | 3
degrees
  device on | 63 [61 to 109]
  device off | 60 [50 to 106]

29. Secondary Outcome: Subjective Benefit for a Control Group: Speech, Spatial, and Qualities of Hearing Scale (SSQ)
Description: Subjects completed subjective questionnaires. For the Speech, Spatial, and Qualities of hearing questionnaire, participants rank their perceived abilities on a scale of 0-10. Higher values indicate more perceived abilities. Results are reported as the average responses across questions for each subscale (Speech Hearing, Spatial Hearing, and Qualities of Hearing). Results are also reported as the total score at each interval, which is the average of the responses from all questions for the questionnaire.
  Participants in the control group had at least 12 months of listening experience with their implanted bone-conduction device prior to study participation.
Time Frame: Assessment completed after 12 months of implantable bone-conduction listening experience
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Control Group: Recipients of a Bone-conduction Device on the Affected Side
Number analyzed (Participants) | 3
score on a scale
  speech hearing subscale | 4.5 [3.7 to 8.6]
  spatial hearing subscale | 1.7 [1.1 to 7.4]
  qualities of hearing subscale | 5.2 [5.0 to 7.7]
  Total score | 3.6 [3.5 to 7.8]

30. Secondary Outcome: Subjective Benefit for a Control Group: Abbreviated Profile of Hearing Aid Benefit (APHAB)
Description: Subjects completed subjective questionnaires. For the Abbreviated Profile of Hearing Aid Benefit, participants rank their perceived difficulty on a scale of 1-99, with lower values indicate less perceived difficulty. Results are reported as the average responses for each of the four subscales: ease of communication, reverberation, effectiveness in background noise, and reverberation. The global score is the average response across questions for the ease of communication, reverberation, and effectiveness in background noise subscales.
  Participants in the control group had at least 12 months of listening experience with their implanted bone-conduction device prior to study participation.
Time Frame: Assessment completed after 12 months of implantable bone-conduction listening experience
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Control Group: Recipients of a Bone-conduction Device on the Affected Side
Number analyzed (Participants) | 3
score on a scale
  global score | 26.3 [12.3 to 45.2]
  ease of communication | 19.2 [12.3 to 60.0]
  reverberation | 39.5 [12.3 to 54.0]
  effectiveness in background noise | 41.7 [12.3 to 62.2]
  aversiveness to sounds | 4.7 [4.7 to 12.3]

31. Other Pre Specified Outcome: Change in Pitch Perception With the Cochlear Implant Over the Post-activation Period
Description: Participants completed an adaptive pitch matching task that compared the pitch of acoustic stimulation presented to their normal hearing ear with the perception of stimulation from the cochlear implant. Two stimuli were used: clicks & tones. Pitch perception was evaluated for the 5 most apical electrodes. A normalized score was obtained (normalized score = geometric mean of the responses / electric center frequency of the evaluated electrode); that is, the normalized score = perceived frequency / frequency information presented by the electrode. Results are reported as the averaged normalized score for clicks & tones for each electrode (electrodes 1-5) at each interval (1, 3, 6, and 12 months post-activation). A value of 1.0 indicates the participant perceived the same frequency as the center frequency presented by the electrode. A value < 1.0 indicates a lower perceived pitch and a value > 1.0 indicates a higher perceived pitch than the electric frequency information.
Time Frame: post-activation period (1, 3, 6, and 12 months post-activation)
Population: 19 of the 20 participants in the single-sided deafness/unilateral hearing loss group elected to complete the pitch matching task on the five most apical electrodes. One participant missed the 1-month and 3-month intervals. Another participant missed the 6-month interval.
Measure: Mean (Standard Deviation); unit: normalized score
Groups:
- Single-sided Deafness/Unilateral Hearing Loss Cohort: participants with a cochlear implant in the affected ear and normal to near-normal hearing in the contralateral ear
Arm/Group | Single-sided Deafness/Unilateral Hearing Loss Cohort
Number analyzed (Participants) | 19
normalized score
  1-month: electrode 1, click: number analyzed (Participants) | 18
  1-month: electrode 1, click | 1.2 (0.4)
  1-month: electrode 1, tone: number analyzed (Participants) | 18
  1-month: electrode 1, tone | 1.3 (0.4)
  1-month: electrode 2, click: number analyzed (Participants) | 18
  1-month: electrode 2, click | 1.0 (0.4)
  1-month: electrode 2, tone: number analyzed (Participants) | 18
  1-month: electrode 2, tone | 1.0 (0.2)
  1-month: electrode 3, click: number analyzed (Participants) | 18
  1-month: electrode 3, click | 0.9 (0.2)
  1-month: electrode 3, tone: number analyzed (Participants) | 18
  1-month: electrode 3, tone | 1.0 (0.4)
  1-month: electrode 4, click: number analyzed (Participants) | 18
  1-month: electrode 4, click | 0.8 (0.2)
  1-month: electrode 4, tone: number analyzed (Participants) | 18
  1-month: electrode 4, tone | 0.9 (0.2)
  1-month: electrode 5, click: number analyzed (Participants) | 17
  1-month: electrode 5, click | 0.9 (0.4)
  1-month: electrode 5, tone: number analyzed (Participants) | 17
  1-month: electrode 5, tone | 0.9 (0.2)
  3-month: electrode 1, click: number analyzed (Participants) | 18
  3-month: electrode 1, click | 1.1 (0.5)
  3-month: electrode 1, tone: number analyzed (Participants) | 18
  3-month: electrode 1, tone | 1.2 (0.3)
  3-month: electrode 2, click: number analyzed (Participants) | 18
  3-month: electrode 2, click | 1.0 (0.4)
  3-month: electrode 2, tone: number analyzed (Participants) | 18
  3-month: electrode 2, tone | 0.9 (0.2)
  3-month: electrode 3, click: number analyzed (Participants) | 18
  3-month: electrode 3, click | 0.8 (0.2)
  3-month: electrode 3, tone: number analyzed (Participants) | 18
  3-month: electrode 3, tone | 0.8 (0.2)
  3-month: electrode 4, click: number analyzed (Participants) | 17
  3-month: electrode 4, click | 0.8 (0.2)
  3-month: electrode 4, tone: number analyzed (Participants) | 17
  3-month: electrode 4, tone | 0.7 (0.2)
  3-month: electrode 5, click: number analyzed (Participants) | 16
  3-month: electrode 5, click | 0.8 (0.3)
  3-month: electrode 5, tone: number analyzed (Participants) | 16
  3-month: electrode 5, tone | 0.7 (0.2)
  6-month: electrode 1, click: number analyzed (Participants) | 18
  6-month: electrode 1, click | 1.2 (0.4)
  6-month: electrode 1, tone: number analyzed (Participants) | 18
  6-month: electrode 1, tone | 1.2 (0.4)
  6-month: electrode 2, click: number analyzed (Participants) | 18
  6-month: electrode 2, click | 1.2 (0.3)
  6-month: electrode 2, tone: number analyzed (Participants) | 18
  6-month: electrode 2, tone | 1.0 (0.3)
  6-month: electrode 3, click: number analyzed (Participants) | 18
  6-month: electrode 3, click | 1.0 (0.4)
  6-month: electrode 3, tone: number analyzed (Participants) | 18
  6-month: electrode 3, tone | 0.9 (0.3)
  6-month: electrode 4, click: number analyzed (Participants) | 17
  6-month: electrode 4, click | 0.9 (0.3)
  6-month: electrode 4, tone: number analyzed (Participants) | 17
  6-month: electrode 4, tone | 0.8 (0.2)
  6-month: electrode 5, click: number analyzed (Participants) | 16
  6-month: electrode 5, click | 0.8 (0.3)
  6-month: electrode 5, tone: number analyzed (Participants) | 16
  6-month: electrode 5, tone | 0.8 (0.2)
  12-month: electrode 1, click | 1.2 (0.4)
  12-month: electrode 1, tone | 1.3 (0.3)
  12-month: electrode 2, click | 1.1 (0.4)
  12-month: electrode 2, tone | 1.1 (0.3)
  12-month: electrode 3, click | 0.9 (0.3)
  12-month: electrode 3, tone | 1.0 (0.3)
  12-month: electrode 4, click: number analyzed (Participants) | 18
  12-month: electrode 4, click | 0.8 (0.2)
  12-month: electrode 4, tone: number analyzed (Participants) | 18
  12-month: electrode 4, tone | 0.9 (0.2)
  12-month: electrode 5, click: number analyzed (Participants) | 16
  12-month: electrode 5, click | 0.9 (0.2)
  12-month: electrode 5, tone: number analyzed (Participants) | 16
  12-month: electrode 5, tone | 0.9 (0.3)
Statistical Analysis 1: Comparison: Single-sided Deafness/Unilateral Hearing Loss Cohort; A linear mixed effects model compared the main effects of target stimulus (click, tone), electrode (1-5), and interval (1, 3, 6, and 12 months) on the normalized pitch match; Test type: Superiority; p < 0.923, Mixed Models Analysis; Main effect: electrode (p<0.001), target stimulus (p=0.923), and interval (p=0.226). Interaction: electrode and interval (p=0.496)
Statistical Analysis 2: Comparison: Single-sided Deafness/Unilateral Hearing Loss Cohort; Correlation between pitch perception (normalized mean pitch match) and word recognition with the CI alone; Test type: Other; p > 0.164, bivariate pearson correlation
Statistical Analysis 3: Comparison: Single-sided Deafness/Unilateral Hearing Loss Cohort; Correlation between pitch perception (normalized mean pitch match) and speech recognition in noise (masker from the front, masker towards the better hearing ear, and masker towards the poorer hearing ear); Test type: Other — bivariate pearson correlation; p > 0.367, bivariate pearson correlation
Statistical Analysis 4: Comparison: Single-sided Deafness/Unilateral Hearing Loss Cohort; Correlation between pitch perception (normalized mean pitch match) and sound source localization (RMS error); Test type: Other — bivariate pearson correlation; p > 0.349, bivariate pearson correlation

32. Post Hoc Outcome: Unaided Hearing in the Implanted Ear Over the Study Period.
Description: The unaided hearing thresholds were measured preoperatively and post-operatively/post-activation. Twenty-five participants with SSD or AHL had an unaided threshold at 125 Hz of 80 dB HL or better. Their unaided thresholds were reviewed with respect to hearing preservation. The data from the SSD and AHL group were combined to review hearing preservation with long arrays. The inclusion criteria for the implanted ear were the same for the SSD and AHL groups and all subjects received the same 31.5 mm electrode array.
Time Frame: pre-operative, initial activation, and post-activation intervals (1, 3, 6, 9, and 12-months).
Population: Participants in the SSD/UHL and AHL groups that presented with an unaided threshold at 125 Hz of 80 dB HL or better (n=25). A value of 100 dB HL was entered for cases of no response.
  Nine participants had a threshold of 95 dB HL or better at initial activation and were reviewed over the post-activation period. Two participants did not complete the 9-month and one participant did not complete the 12-month.
Measure: Mean (Standard Deviation); unit: decibel hearing level
Groups:
- Single-sided Deafness/Unilateral Hearing Loss and Asymmetric Hearing Loss Groups Combined: The data from both groups (SSD and AHL) were combined.
Arm/Group | Single-sided Deafness/Unilateral Hearing Loss and Asymmetric Hearing Loss Groups Combined
Number analyzed (Participants) | 25
decibel hearing level
  preoperative | 62 (16)
  initial activation | 93 (13)
  1-month post-activation: number analyzed (Participants) | 9
  1-month post-activation | 76 (18)
  3-month post-activation: number analyzed (Participants) | 9
  3-month post-activation | 69 (10)
  6-month post-activation: number analyzed (Participants) | 9
  6-month post-activation | 76 (14)
  9-month post-activation: number analyzed (Participants) | 9
  9-month post-activation | 73 (15)
  12-month post-activation: number analyzed (Participants) | 9
  12-month post-activation | 74 (14)
Statistical Analysis 1: Comparison: Single-sided Deafness/Unilateral Hearing Loss and Asymmetric Hearing Loss Groups Combined; Comparison of the unaided threshold at 125 Hz at the preoperative and initial activation intervals for the 25 participants with unaided threshold of 80 dB HL or better at the preoperative interval. The data from the SSD and AHL group were combined to review hearing preservation with long arrays. The inclusion criteria for the implanted ear were the same for the SSD and AHL groups and all subjects received the same 31.5 mm electrode array; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Single-sided Deafness/Unilateral Hearing Loss and Asymmetric Hearing Loss Groups Combined; Comparison of the unaided threshold at 125 Hz from the initial activation to the 12-month post-activation interval for the 9 participants with an unaided threshold of 95 dB HL or better at the initial activation interval. The data from the SSD and AHL group were combined to review hearing preservation with long arrays. The inclusion criteria for the implanted ear were the same for the SSD and AHL groups and all subjects received the same 31.5 mm electrode array; Test type: Superiority; p = 0.47, ANOVA; generalized linear mixed-effects model

33. Post Hoc Outcome: Localization With a Bone-conduction Device Over Time, Measured in Root-mean-squared (RMS) Error
Description: Subjects were asked to identify the noise source from an 11-speaker array. The intensity level of the stimulus was randomly varied (10 dB around 70 dB SPL) to limit the listener relying on level effects. Responses at each intensity level (i.e., 60, 70, and 80 dB SPL) for a given sound source (speaker) were combined. Performance was measured with a bone conduction device preoperatively and 12 months post-activation. Overall root-mean-square (RMS) error is the difference between the sound source azimuth and the response azimuth and a lower score indicates more accurate localization of the sound source.
Time Frame: preoperative and 12-month intervals
Population: Three participants in the asymmetric hearing loss group did not complete the task at the 12-month interval.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
degrees
  preoperative | 70 (19) | 76 (18)
  12-month: number analyzed (Participants) | 20 | 17
  12-month | 69 (19) | 80 (14)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; A paired samples t-test compared the performance with the bone-conduction device at the preoperative and 12-month intervals; Test type: Superiority; p = 0.739, t-test, 2 sided
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 33, analysis 1]; Test type: Superiority; p = 0.553, t-test, 2 sided

34. Post Hoc Outcome: Speech Recognition in Noise With a Bone-conduction Device Over Time, Measured With AzBio Sentences
Description: Speech recognition with a bone-conduction device was compared at the preoperative and 12-month intervals. Performance was evaluated for the AzBio sentences in a 10-talker masker (0 dB SNR) presented with the target and masker from the front, the target from the front and masker to the acoustic hearing, and target from the front and masker towards the affected ear.
Time Frame: preoperative and 12-month intervals
Population: Thirteen participants with asymmetric hearing loss completed the task at the preoperative and 12-month intervals at 0 dB SNR.
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
percent correct
  preoperative, speech front and noise front: number analyzed (Participants) | 20 | 13
  preoperative, speech front and noise front | 32 (17) | 17 (12)
  preoperative, speech front and noise to the acoustic ear: number analyzed (Participants) | 20 | 13
  preoperative, speech front and noise to the acoustic ear | 18 (18) | 6 (8)
  preoperative, speech front and noise to the affected ear: number analyzed (Participants) | 20 | 13
  preoperative, speech front and noise to the affected ear | 61 (28) | 24 (18)
  12-month, speech front and noise front: number analyzed (Participants) | 20 | 13
  12-month, speech front and noise front | 42 (16) | 16 (12)
  12-month, speech front and noise to the acoustic ear: number analyzed (Participants) | 20 | 13
  12-month, speech front and noise to the acoustic ear | 29 (18) | 1 (3)
  12-month, speech front and noise to the affected ear: number analyzed (Participants) | 20 | 13
  12-month, speech front and noise to the affected ear | 69 (18) | 31 (20)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; A repeated-measures ANOVA assessed the effects of interval (preoperative and 12-months) and masker condition (front, acoustic ear, or affected ear) on performance with the bone conduction device; Test type: Superiority; p < 0.345, ANOVA — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis; Main effect: interval (p=0.027) and masker condition (p<0.001). Interaction: interval and masker condition (p=0.345)
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 34, analysis 1]; Test type: Superiority; p < 0.577, ANOVA — Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis; Main effect: masker condition (p<0.001) and interval (p=0.577). Interaction: interval and masker condition (p=0.055)

35. Post Hoc Outcome: Pitch Perception on 5 Most Apical Electrodes With the Fine Structure Coding Strategy (FS4) Versus the Continuous Interleaved Sampling (CIS) Coding Strategy
Description: 9 participants repeated the pitch perception task at the 12-month interval while listening to the CIS strategy. FS4 & CIS strategies differ in whether or not fine structure cues are provided on the 4 most apical electrodes; there is no difference in the cues provided by electrode 5. An adaptive task compared the pitch of acoustic stimulation presented to the normal hearing ear with the stimulation from the cochlear implant. A normalized score was obtained (normalized score = geometric mean of the responses / electric center frequency of the evaluated electrode); that is, the normalized score = perceived frequency / presented frequency information. Results are reported as the averaged normalized score for clicks & tones for each electrode. A value of 1.0 indicates the perceived frequency was the same as the electric frequency information. A value < 1.0 indicates a lower perceived pitch and a value > 1.0 indicates a higher perceived pitch than the electric frequency information.
Time Frame: 12-month interval
Population: One participant did not complete testing for electrode 5
Measure: Mean (Standard Deviation); unit: normalized score
Arm/Group | Single-sided Deafness/Unilateral Hearing Loss Cohort
Number analyzed (Participants) | 9
normalized score
  electrode 1, FS4 | 1.2 (0.3)
  electrode 1, CIS | 1.5 (0.3)
  electrode 2, FS4 | 1.0 (0.2)
  electrode 2, CIS | 1.1 (0.3)
  electrode 3, FS4 | 0.9 (0.2)
  electrode 3, CIS | 0.9 (0.2)
  electrode 4, FS4 | 0.9 (0.3)
  electrode 4, CIS | 0.8 (0.3)
  electrode 5, FS4: number analyzed (Participants) | 8
  electrode 5, FS4 | 0.9 (0.2)
  electrode 5, CIS: number analyzed (Participants) | 8
  electrode 5, CIS | 0.9 (0.2)
Statistical Analysis 1: Comparison: Single-sided Deafness/Unilateral Hearing Loss Cohort; A linear mixed effect model assessed the main effects of stimulus, electrode, and coding strategy, and their interactions; Test type: Superiority; p > 0.023, Mixed Models Analysis; Main effect: coding strategy (p=0.023). Interaction: coding strategy and electrode (p=0.044). All other main effects and interactions were p>0.160
Statistical Analysis 2: Comparison: Single-sided Deafness/Unilateral Hearing Loss Cohort; Paired samples t-tests evaluated whether pitch perception (mean normalized pitch) differed between coding strategy for each electrode; Test type: Superiority; p > 0.035, t-test, 2 sided; Pitch perception for electrode 1 (p=0.035). All other comparisons were p>0.318

36. Post Hoc Outcome: Localization in the Unaided Condition and With a Bone-conduction Device, Measured in Root-mean-squared Error.
Description: Subjects were asked to identify the noise source from an 11-speaker array with a bone-conductive device on versus off. The intensity level of the stimulus was randomly varied (10 dB around 70 dB SPL) to limit the listener relying on level effects. Responses at each intensity level (i.e., 60, 70, and 80 dB SPL) for a given sound source (speaker) were combined. Results are reported in root-mean-squared (RMS) error. A lower value indicates better performance. Results are compared at the preoperative and 12-month post-activation intervals.
Time Frame: preoperative and 12-month post-activation intervals.
Population: One participant in the asymmetric group withdrew before the 12-month interval. Two additional participants in the asymmetric hearing loss group did not complete the procedure with the bone-conduction device at the 12-month interval.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
degrees
  before surgery, unaided | 66 (20) | 76 (19)
  before surgery, bone conduction device | 70 (19) | 76 (18)
  12-month, unaided: number analyzed (Participants) | 20 | 19
  12-month, unaided | 68 (18) | 79 (17)
  12-month, bone conduction device: number analyzed (Participants) | 20 | 17
  12-month, bone conduction device | 69 (19) | 80 (14)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; A repeated-measures ANOVA assessed the effects of condition (unaided, bone-conduction device) and interval (preoperative, 12-month) and their interaction on sound source localization; Test type: Superiority; p > 0.084, ANOVA; Main effects: condition (p=0.960) and interval (p=0.084). Interaction: condition and interval (p=0.433)
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 36, analysis 1]; Test type: Superiority; p > 0.434, ANOVA; Main effect: condition (p=0.434) or interval (p=0.687). Interaction: condition and interval (p=0.678)

37. Post Hoc Outcome: Speech Recognition in Noise in the Unaided Condition and With a Bone-conduction Device, Measured With AzBio Sentences
Description: Speech recognition in noise with the AzBio sentences in 3 masker conditions (masker from the front, masker towards the better hearing ear, and masker towards the poorer hearing ear) at the preoperative and 12-month intervals in the unaided condition and with a bone-conduction device. Percent correct results were converted to rationalized arcsine units (RAUs) which helps to control for floor and ceiling effects in the perception correct data (e.g., <20% correct).
Time Frame: preoperative interval and 12-month post-activation interval.
Population: All participants in the UHL/SSD group completed the task at 0 dB SNR. Not all participants in the AHL group completed the task at 0 dB SNR.
Measure: Mean (Standard Deviation); unit: rationalized arcsine units
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group
Number analyzed (Participants) | 20 | 20
rationalized arcsine units
  preop, unaided, masker towards better ear: number analyzed (Participants) | 20 | 13
  preop, unaided, masker towards better ear | 11 (21) | -13 (12)
  preop, bone-conduction, masker towards better ear: number analyzed (Participants) | 20 | 13
  preop, bone-conduction, masker towards better ear | 11 (26) | -5 (16)
  12-month, unaided, masker towards better ear: number analyzed (Participants) | 20 | 15
  12-month, unaided, masker towards better ear | 18 (23) | -14 (16)
  12-month, bone-conduction, masker towards better ear: number analyzed (Participants) | 20 | 13
  12-month, bone-conduction, masker towards better ear | 28 (20) | -18 (9)
  preop, unaided, masker from front: number analyzed (Participants) | 20 | 13
  preop, unaided, masker from front | 38 (11) | 14 (17)
  preop, bone-conduction, masker from front: number analyzed (Participants) | 20 | 13
  preop, bone-conduction, masker from front | 29 (22) | 13 (18)
  12-month, unaided, masker from front: number analyzed (Participants) | 20 | 15
  12-month, unaided, masker from front | 42 (11) | 20 (18)
  12-month, bone-conduction, masker from front: number analyzed (Participants) | 20 | 13
  12-month, bone-conduction, masker from front | 42 (17) | 12 (20)
  preop, unaided, masker towards poorer ear: number analyzed (Participants) | 20 | 13
  preop, unaided, masker towards poorer ear | 85 (12) | 40 (18)
  preop, bone-conduction, masker towards poorer ear: number analyzed (Participants) | 20 | 13
  preop, bone-conduction, masker towards poorer ear | 61 (33) | 22 (22)
  12-month, unaided, masker towards poorerear: number analyzed (Participants) | 20 | 15
  12-month, unaided, masker towards poorerear | 86 (15) | 37 (26)
  12-month, bone-conduction, masker from towards poorer ear: number analyzed (Participants) | 20 | 13
  12-month, bone-conduction, masker from towards poorer ear | 70 (10) | 29 (24)
Statistical Analysis 1: Comparison: Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group; A repeated-measures ANOVA assessed the effects of condition (unaided, bone-conduction device), interval (preoperative, 12-month), and masker condition and their 2-way and 3-way interactions on speech recognition in noise; Test type: Superiority; p < 0.935, ANOVA — Percent correct converted to rationalized arcsine units (RAU) prior to analysis; Main effects: condition (p=0.018), interval (p=0.012), and masker (p<0.001). Interactions: interval and masker (p<0.001). Other interactions: p>0.117
Statistical Analysis 2: Comparison: Cochlear Implant: Asymmetric Hearing Loss Group; [analysis description as in outcome 37, analysis 1]; Test type: Superiority; p < 0.977, ANOVA — A Greenhouse-Geisser correction was applied as indicated by the Mauchly test of sphericity; Effects: interval (p=0.012) and masker (p<0.001). Interactions: interval&masker (p=0.020) & condition, interval, &masker (p=0.035). Others: (p>0.131)

ADVERSE EVENTS:
Time Frame: 12 months post-activation
Groups:
- Control Group (Recipients of a Bone-conduction Device): Recipients of a bone-conduction device (alternative treatment technology) with at least 12 months of device use.
Arm/Group | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group | Cochlear Implant: Asymmetric Hearing Loss Group | Control Group (Recipients of a Bone-conduction Device)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/3
Other Adverse Events (participants affected / at risk) | 8/20 | 5/20 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cochlear Implant: Unilateral Hearing Loss/Single-sided Hearing Loss Group (N=20) | Cochlear Implant: Asymmetric Hearing Loss Group (N=20) | Control Group (Recipients of a Bone-conduction Device) (N=3)
vertigo / dizziness (Ear and labyrinth disorders) | 5 | 1 | 0
light-headedness & nausea (Ear and labyrinth disorders) | 1 | 0 | 0
imbalance (Ear and labyrinth disorders) | 0 | 1 | 0
nystagmus (Ear and labyrinth disorders) | 1 | 0 | 0
drainage (General disorders) | 0 | 1 | 0
headache (General disorders) | 0 | 1 | 0
facial stimulation (General disorders) | 0 | 1 | 0
bleeding at surgical site (General disorders) | 1 | 0 | 0
short circuit (Product Issues) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Unable to reach maximum enrollment in the control group (bone conduction device users).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT02203305/Prot_SAP_000.pdf